# Statistical Analysis Plan: Work2Prevent - Phase 2

**PROTOCOL:** ATN 151: Work2Prevent: Employment as HIV prevention

for young men who have sex with men (YMSM) and young

transgender women (YTW)

PROTOCOL DATE: May 23, 2017

Revised August 5, 2019

**PROTOCOL VERSION:** 5.2

CLINICALTRIALS.GOV ID: NCT03313310

**SPONSOR:** The Eunice Kennedy Shriver National Institute of Child

Health and Human Development (NICHD)

with co-funding from:

National Institute on Drug Abuse (NIDA),

National Institute of Mental Health (NIMH), and National Institute on Minority Health and Health

Disparities (NIMHD)

SAP DATE: December 13, 2019

SAP VERSION: 2.0

SAP PREPARED BY: ATN Coordinating Center

**Collaborative Studies Coordinating Center** 

**Department of Biostatistics** 

The University of North Carolina at Chapel Hill 123 W. Franklin Street, Suite 450, CB# 8030

Chapel Hill, NC 27599-8030

AUTHORS: Myra A. Carpenter, PhD

Micah McCumber, MS Cara M. Nordberg, MPH Justin Demonte, BS Betty Rupp, MPH

# SIGNATURE PAGE

| Name | Role | Signature | Date |
|----------------|------------------------|-----------|------|
| Lisa Strader | ATN CC Co-Investigator | | |
| Brandon Hill | Principal Investigator | | |
| Darnell Motley | Site Investigator | | |

# **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 7 |
|----|-------------------------------------------------------------------|-----|
| | 1.1. OBJECTIVES AND RESEARCH HYPOTHESES | 7 |
| 2. | STUDY METHODS | . 7 |
| | 2.1. Study Design | 7 |
| | 2.2. Study Population | 7 |
| | 2.3. Sample Size Information | 8 |
| 3. | ANALYSIS POPULATIONS | . 8 |
| | 3.1. PER PROTOCOL POPULATION | 9 |
| 4. | STUDY ASSESSMENTS | 9 |
| | 4.1. Primary Outcomes | 9 |
| | 4.1.1. Information Systems Success Model Score (T2) | 9 |
| | 4.1.2. Workshop Completion (T2) | 9 |
| | 4.1.3. Change in Job-Seeking Self-Efficacy Scale Score (T1 to T3) | 10 |
| | 4.1.4. Change in Protean Career Attitudes Scale Score (T1 to T3) | 10 |
| | 4.2. SECONDARY OUTCOMES | 10 |
| | 4.2.1. Change in Self-Reported Hours Worked Per Week (T1 to T3) | 10 |
| | 4.2.2. Change in Self-Reported Sexual Risk Behaviors (T1 to T3) | 10 |
| | 4.2.3. Change in Chlamydia Test Result (T1 to T3) | 11 |
| | 4.2.4. Change in Gonorrhea Test Result (T1 to T3) | 11 |
| | 4.2.5. Reactive HIV Test (T3) | 11 |
| 5. | STATISTICAL ANALYSIS | 11 |
| | 5.1. GENERAL CONSIDERATIONS | 11 |
| | 5.2. MISSING DATA | 12 |
| | 5.3. Subject Disposition Analyses | 12 |
| | 5.4. Analysis of Primary Outcomes | 12 |
| | 5.5. Analysis of Secondary Outcomes | 12 |
| | 5.6. ANALYSIS OF SAFETY EVENTS | 12 |
| RE | FERENCES | 14 |
| ΑP | PENDIX | 15 |
| 1. | PRIMARY OUTCOMES | 15 |

| | 1.1. INFORMATION SYSTEMS SUCCESS MODEL (ISSM) SCALE | 15 |
|---|---|---|
| | 1.1.1. ISSM Subscale 1: Information Quality (IQ) Score | 15 |
| | 1.1.2. ISSM Subscale 2: Handbook Quality (HQ) Score | 15 |
| | 1.1.3. ISSM Subscale 3: Perceived Usefulness (PU) Score | 16 |
| | 1.1.4. ISSM Subscale 4: Overall Score | 16 |
| | 1.1.5. Information Systems Success Model (ISSM) Score | 17 |
| | 1.2. WORKSHOP COMPLETION | 17 |
| | 1.2.1. Number of Workshops Attended | 17 |
| | 1.2.2. Workshop Completion | 17 |
| | 1.3. JOB SEEKING SELF-EFFICACY SCALE SCORE | 18 |
| | 1.3.1. Job Seeking Self-Efficacy Score at Baseline (T1) | 18 |
| | 1.3.2. Job Seeking Self-Efficacy Score at Post-Intervention (T2) | 18 |
| | 1.3.3. Job Seeking Self-Efficacy Score at Month 8 Follow-Up (T3) | 19 |
| | 1.3.4. Change in Job Seeking Self-Efficacy Score from Baseline to Month 8 Follow (T1T3) | - |
| | 1.4. PROTEAN CAREER ATTITUDES SCALE (PCA) SCORE: | 20 |
| | 1.4.1. PCA Subscale 1: Self-Directed Attitudes Scale Score | 20 |
| | 1.4.2. PCA Subscale 2: Values-Driven Attitudes Scale Score | 21 |
| | 1.4.3. Scale: Protean Career Attitudes (PCA) Scale | 22 |
| 2. | SECONDARY OUTCOMES | 24 |
| | 2.1. SELF-REPORTED EMPLOYMENT | 24 |
| | 2.1.1. Change in Self-Reported Hours Worked Per Week from Baseline to Month Follow-Up (T1T3) | |
| | 2.2. SELF-REPORTED SEXUAL RISK BEHAVIORS | 24 |
| | 2.2.1. Self-Reported Sexual Risk Behavior at Baseline (T1) | 24 |
| | 2.2.2. Self-Reported Sexual Risk Behavior at Baseline (T3) | 25 |
| | 2.2.3. Change in Self-Reported Risk Behavior from Baseline to Month 8 Follow-U | |
| | 2.3. CHLAMYDIA INFECTIONS: | 25 |
| | 2.3.1. Chlamydia Result at Baseline (T1) | 25 |
| | 2.3.2. Chlamydia Result at Month 8 Follow-Up (T3) | |
| | 2.3.3. Change in Chlamydia Result from Baseline to Month 8 Follow-Up (T1T3) | 28 |

| 2.4. GONORRHEA INFECTIONS: | 29 |
|---|---|
| 2.4.1. Gonorrhea Result at Baseline (T1) | 29 |
| 2.4.2. Gonorrhea Result at Month 8 Follow-Up (T3) | 30 |
| 2.4.3. Change in Gonorrhea Result from Baseline to Month 8 Follow-Up (T1T3) | 32 |
| 2.5. REACTIVE HIV TEST | 33 |

#### LIST OF ABBREVIATIONS

AIDS Acquired Immunodeficiency Syndrome

ATN Adolescent Medicine Trials Network for HIV/AIDS Interventions

CAI Condomless Anal Intercourse CC ATN Coordinating Center

CSCC Collaborative Studies Coordinating Center

HIV Human Immunodeficiency Virus

HQ Handbook Quality IQ Information Quality

ISSM Information Systems Success Model

JSS Job-Seeking Self-Efficacy
MSM Men who have Sex with Men

NICHD Eunice Kennedy Shriver National Institute of Child Health and Human Development

NIDA National Institute on Drug Abuse
NIMH National Institute of Mental Health

NIMHD National Institute on Minority Health and Health Disparities

PCA Protean Career Attitudes
PU Perceived Usefulness
SDA Self-Directed Attitudes

STI Sexually Transmitted Infection

T1 Baseline Visit

T2 Post-Intervention Visit at 0-2 weeks post-intervention T3 Follow-up at 8-months (±4 weeks) post-intervention

VDA Values-Driven Attitudes

W2P Work2Prevent

YMSM Young Men who have Sex with Men

YTW Young Transgender Women

#### 1. INTRODUCTION

Work2Prevent (W2P) is a project designed to adapt, tailor, and pilot-test a novel social and structural-level HIV intervention for Young Men who have Sex with Men (YMSM) and Young Transgender Women (YTW) of color aimed at increasing economic stability (i.e., employment) through youth empowerment and asset development, and decreasing HIV risk behaviors (i.e., sex work) associated with social and economic marginalization. This document gives details of the planned statistical analysis for Phase 2 of the intervention.

## 1.1. Objectives and Research Hypotheses

The primary objective of Phase 2 is to pilot-test the intervention among up to 70 at-risk YMSM and YTW of color in order to evaluate feasibility and acceptability. Investigators hypothesize the intervention will increase job self-efficacy and readiness, as well as decrease HIV risk behaviors and STI and HIV infections.

#### 2. STUDY METHODS

## 2.1. Study Design

W2P is a single-arm longitudinal pre and post study of the social and structural-level employment intervention to evaluate feasibility, acceptability, and satisfaction of the intervention program, and preliminary efficacy for study outcomes assessed at Baseline (T1), Post-Intervention (T2, 0 to 2 weeks post workshop completion), and 8-Month Follow-up (±4 weeks) (T3). The study employment intervention is comprised of four structured workshops presented over a 2-week period.

The study aims to enroll up to 70 at-risk YMSM and YTW of color over a 6-month period. The intervention workshops will be completed within 12 weeks of enrollment. Each participant will then be assessed 8-months (±4 weeks) post-intervention.

Study outcomes include: (1) Job self-efficacy and readiness; (2) HIV risk behaviors; (3) Employment; and (4) STI and HIV infections.

### 2.2. Study Population

All intervention study participants are Black or African American or Hispanic or Latinos males, including transgender women (those assigned male at birth), ages 16-24, who identify as either an (1) MSM or gay or bisexual man or as a (2) transgender woman or transsexual male-to-female or transwoman.

## Participant Inclusion Criteria<sup>1</sup>:

- 1. Being male or assigned male at birth (YTW)
- 2. Identifying as YMSM or gay bisexual man or transgender woman or transwoman
- 3. Identifying as African American or Black, Hispanic or Latino, or as a racial or ethnic minority or person of color
- 4. 16-24 years old
- 5. English-speaking (primary)
- 6. HIV negative or of unknown status
- 7. Currently unemployed but seeking employment, or employed only part-time (average of 35 hours or less per week)
- 8. Able to attend a 4-session employment program

### Participant Exclusion Criteria:

- 1. Individuals identifying as non-Hispanic white
- 2. Individuals not assigned male at birth

#### 2.3. Sample Size Information

This study aims to enroll up to 70 participants with at least 50 of these participants completing the study ( $\sim$ 70% retention rate). Given the exploratory nature of this study and limited access to this population, a power calculation was not performed. A repeated measures design was chosen to reduce the variability in the estimate of the treatment effect, at the expense of having a comparison group. In addition, practice or fatigue effects from repetition may affect certain outcomes (e.g. protean career attitudes scale and subscales). This trade-off was appropriate given the exploratory nature of a pilot study and the limited access to the study population.

## 3. ANALYSIS POPULATIONS

Only participants who are enrolled at Baseline (complete the T1 survey) will be included in the primary and secondary analyses. Screen-failures will not be included in these analyses.

### 3.1. Intent-to-Treat Population

All participants who completed T3 will be included in intent-to-treat analyses involving variables measuring changes from T1 to T3 (see sections 4.1.3-4.1.4 and 4.2.1-4.2.5 below).

All participants who completed at least one workshop will be included in intent-to-treat analyses involving workshop evaluation and workshop completion variables (see sections 4.1.1,

<sup>&</sup>lt;sup>1</sup> The original inclusion criteria included "Considered 'at-risk' for HIV based on 6-item risk assessment". The removal of this criterion was approved on August 16, 2018 as part of protocol v4.0 and eligibility was rerun retrospectively for those who completed the Screener Survey (SCR) prior to the inclusion criteria modification.

4.1.2 below). This population will form the basis for both the primary and secondary analyses of the efficacy and safety endpoints.

#### 3.2. Per Protocol Population

Youth who attend at least two of the four planned intervention workshops and complete T3 will comprise the per protocol population. This population will form the basis for both the primary and secondary supportive analyses of the efficacy and safety endpoints.

#### 4. STUDY ASSESSMENTS

| | | Baseline | Post- | 8-Month |
|---|---|---|---|---|
| Study Assessments | Pre-Screening | (T1) | Intervention (T2) | Follow-Up (T3) |
| Screener Questionnaire (SCR) | X | | | |
| Eligibility Form (ELG) | | Χ | | |
| Baseline Questionnaire (BSL) | | Χ | | |
| Biospecimen Collection Form (BIC) | | Х | | Х |
| Biospecimen Lab Results<br>Form (BLR) | | Х | | X |
| Workshop Tracking (WTI) | | | X | |
| Workshop Evaluation (EVL) | | | X | |
| Exit Visit Questionnaire (EXQ) | | | | X |

## 4.1. Primary Outcomes

### 4.1.1. Information Systems Success Model Score (T2)

The Information Systems Success Model (ISSM) will be used to assess for intervention acceptability and satisfaction. The 21-item scale measures four sub-domains: information quality, handbook quality, perceived usefulness, and overall satisfaction. Every item is scored on a 1 to 5 scale, with 1 being "Strongly Disagree" and 5 being "Strongly Agree". Responses are averaged within each sub-domain to produce four sub-domain scores. The four sub-domain scores are then averaged to produce an overall ISSM score (range: 1 to 5; higher scores indicate higher acceptability/satisfaction). This scale has been adapted from Horvath et al.<sup>1</sup>

### 4.1.2. Workshop Completion (T2)

Workshop completion will be used to assess for intervention feasibility. The outcome of intervention completion will be defined as having attended at least two of the four workshop sessions and will be measured by tracking participant attendance. Workshop completion may also be defined as the number of workshop sessions attended for use in exploratory analyses.

## 4.1.3. Change in Job-Seeking Self-Efficacy Scale Score (T1 to T3)

Job seeking self-efficacy is defined as one's perceived ability and confidence to perform job search and application activities. The 12-item Job Seeking Self-Efficacy (JSS) scale by Barlow et al<sup>2</sup> uses response values on a 1 to 10 score, with 1 being "Not At All Confident" and 10 being "Very Confident". Reponses are averaged to yield a total score, with higher scores indicating higher self-efficacy. Change in JSS will be calculated by subtracting the JSS score at baseline (T1) from the JSS score at the 8-month follow-up (T3) (range: -9 to +9; negative change indicates decreased self-efficacy, while positive change indicates increased self-efficacy).

## 4.1.4. Change in Protean Career Attitudes Scale Score (T1 to T3)

Protean career attitudes (PCAs) are defined as having self-direction in the pursuit of success in one's work. PCAs have previously been found to be associated with positive career satisfaction and self-perceived success.<sup>3</sup> The validated 7-item scale by Porter et al<sup>4</sup> measures two subdomains: self-directed attitudes and values-driven attitudes. Every item is scored on a 1 to 5 scale, with 1 being "Strongly Disagree" and 5 being "Strongly Agree". Responses are averaged within each sub-domain to produce two sub-domain scores, which are then averaged as well to produce an overall PCA score. Change in PCA score will be calculated by subtracting the score at baseline (T1) from the score at the 8-month follow-up (T3) (range: -4 to +4; negative change indicates decreased PCAs, while positive change indicates increased PCAs).

## 4.2. Secondary Outcomes

## 4.2.1. Change in Self-Reported Hours Worked Per Week (T1 to T3)

Hours worked per week will be self-reported at baseline and at the 8-month follow-up visit as any value between 0 and 99. Change in hours worked per week will be calculated by subtracting the baseline (T1) value from the 8-month follow-up (T3) value. Negative change indicates fewer hours worked per week, while positive change indicates more hours work per week.

### 4.2.2. Change in Self-Reported Sexual Risk Behaviors (T1 to T3)

Sexual risk behaviors will be measured using six yes or no (1 or 0) items assessing for engagement in the following behaviors during the 6 months prior to baseline (T1) and 8-month follow-up (T3) assessments:

- 1. condomless anal intercourse (CAI) with male partner of unknown HIV status
- 2. anal intercourse with ≥3 males
- 3. sex with male partner with a Sexually Transmitted Infection (STI)
- 4. CAI with HIV+ male partner
- 5. anal intercourse with condom failure
- 6. transactional sex work involvement

Responses will be averaged at each assessment. Change in sexual risk behaviors will be calculated by subtracting the average at baseline from the average at the 8-month follow-up (range: -1 to +1; negative change indicates fewer sexual risk behaviors, while positive change indicates more sexual risk behaviors).

## 4.2.3. Change in Chlamydia Test Result (T1 to T3)

Chlamydia infections will be assessed at baseline and 8-month follow up using oral, anal, and urine samples. Each of the three tests yields a positive (1) or negative (0) result. Change in test result will be calculated by subtracting the baseline result from the 8-month follow-up result. Oral, anal, and urine tests will be treated as separate outcomes.

## 4.2.4. Change in Gonorrhea Test Result (T1 to T3)

Gonorrhea infections will be assessed at baseline and 8-month follow up using oral, anal, and urine samples. Each of the three tests yields a positive (1) or negative (0) result. Change in test result will be calculated by subtracting the baseline result from the 8-month follow-up result. Oral, anal, and urine tests will be treated as separate outcomes.

## 4.2.5. Reactive HIV Test (T3)

Testing for HIV will be assessed at baseline and 8-month follow up. The test yields a reactive (1) or non-reactive (0) result. The outcome for reactive HIV test will use the T3 test result.

#### 5. STATISTICAL ANALYSIS

#### 5.1. General Considerations

The analytic plan is designed to determine preliminary efficacy of the intervention by comparing pre/post assessments of employment and sexual risk behaviors. Descriptive statistics will be used to analyze the proportions and central tendencies for participant sociodemographic covariates collected in the surveys. We will first generate frequencies, means, and other measures of central tendency as appropriate to describe our sample and outcomes at each of the three time points (baseline, post-intervention, and 8-month follow-up).

Changes in primary and secondary outcomes between baseline and 8-month follow-up will be assessed using paired t-tests for continuous variables and McNemar's test for matched categorical variables. We will use standard diagnostic tools to assess the appropriateness of the normality assumption (e.g., QQ-plots) and, if approximate normality of the residuals is not tenable, a non-parametric test for continuous paired data, i.e. Wilcoxon sign rank test will be used. All hypothesis testing will be done at an alpha-level of 0.1, given the exploratory nature of the study.

### 5.2. Missing Data

Missing responses to survey questions will be ignored and non-missing data will be used to compute the primary and secondary outcomes. If all components for an outcome are missing, then the outcome will be considered missing. For those outcomes with unique missing data rules, the handling of missing data for each individual outcome are described in the appendix. Missing data patterns will be explored prior to the analysis of the primary and secondary outcomes.

## **5.3. Subject Disposition Analyses**

Number of participants pre-screened, screened, eligible, discontinued, and included in the Per Protocol analysis population will be reported. In addition, the number of participants completing each visit (T1, T2 and T3) and the reasons for patient discontinuation will be tabulated.

## **5.4. Analysis of Primary Outcomes**

Primary outcomes for analyses include Information Systems Success Model score, workshop completion, change in Job-Seeking Self Efficacy Scale score, Protean Career Attitudes Scale score, change in Self-Directed Attitudes Scale score, and change in Values-Driven Attitudes Scale score. Details about these outcomes are described in Section 4.1.

Univariate analyses will be performed as described in Section 5.1. To the extent that data allows, multivariable analyses will adjust for sociodemographic characteristics, workshop attendance, baseline employment status, and study completeness. Analytical models will include linear regression or generalized linear models for continuous outcomes and logistic regression for binary and categorical outcomes.

## 5.5. Analysis of Secondary Outcomes

Secondary outcomes for analyses include change in self-reported hours worked per week, change in self-reported sexual risk behavior, change in chlamydia test results, change in gonorrhea test results, and reactive HIV test result. Details about these outcomes are described in Section 4.2.

Univariate analyses will be performed as described in Section 5.1. Multivariable analyses will adjust for sociodemographic characteristics, workshop attendance, baseline employment status, and study completeness. Analytical models will include linear regression or generalized linear models for continuous outcomes and logistic regression for binary and categorical outcomes.

### 5.6. Analysis of Safety Events

Safety Events will be recorded for participants as needed throughout the study. The number of participants experiencing each safety event will be summarized by severity grade, relationship

to study, and action taken. All safety events will be provided in the safety events data listing. Withdrawals due to safety events will also be reported.

#### REFERENCES

- 1. Horvath KJ, Oakes MJ, Rosser SBR, Danilenko G, Vezina H, Amico RK, Williams ML, Simoni J. Feasibility, Acceptability and Preliminary Efficacy of an Online Peer-to-Peer Social Support ART Adherence Intervention. AIDS Behav., 2013; 17:2031-2044.
- 2. Barlow J, Wright C, Cullen L. *A job-seeking self-efficacy scale for people with physical disabilities: preliminary development and psychometric testing.* Br J Guid Counc., 2002; 30:1, 37-53.
- 3. Volmer J, Spurk D. *Protean and boundaryless career attitudes: relationships with subjective and objective career success.* J Labor Mark Res., 2011; 43:207-218.
- 4. Porter C, Woo SE, Tak J. *Developing and Validating Short Form Protean and Boundaryless Career Attitudes Scales*. J Career Assess., 2016; 24(1):162-181.

### 1. PRIMARY OUTCOMES

### 1.1. INFORMATION SYSTEMS SUCCESS MODEL (ISSM) SCALE

The Information Systems Success Model (ISSM) scale has been adapted from Horvath et al. 2013 to assess intervention acceptability and satisfaction. The scale evaluates four sub-domains: information quality, system quality, perceived usefulness, and overall satisfaction. For each of the calculated scores, higher values indicate better participant-assessed quality.

## 1.1.1. ISSM Subscale 1: Information Quality (IQ) Score

<u>Description</u>: Information Quality is a 6-item sub-scale measured at time point T2 (post-intervention)

to evaluate ease of comprehension, credibility, clarity, and accuracy of the information provided through the intervention using responses to items 7a through 7e and 8a in the Evaluation (EVL) Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4 points, and

5/Strongly Agree = 5 points.

Variable: IQ\_T2\_1

Label: Information Quality Score at T2

Type: Numeric; Range = 1 to 5

<u>Algorithm:</u> IQ\_T2\_1 = MEAN (EVL7a, EVL7b, EVL7c, EVL7d, EVL7e, EVL8a)

If all responses are missing, then then IQ\_T2\_1=Missing. Otherwise, consider mean of

non-missing responses.

### 1.1.2. ISSM Subscale 2: Handbook Quality (HQ) Score

<u>Description</u>: Handbook Quality is a 6-item sub-scale measured at time point T2 (post-intervention) to

evaluate user friendliness and appeal of the workshop handbook provided through the

intervention using responses to items 8b through 8e, 9a, and 9b in the EVL

Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4 points, and 5/Strongly

Agree = 5 points.

Variable: HQ\_T2\_1

Label: Handbook Quality Score at T2

Type: Numeric; Range = 1 to 5

Algorithm: HQ\_T2\_1 = MEAN (EVL8b, EVL8c, EVL8d, EVL8e, EVL9a, EVL9b)

If all responses are missing, then HQ\_T2\_1=Missing. Otherwise, consider mean of non-missing responses.

## 1.1.3. ISSM Subscale 3: Perceived Usefulness (PU) Score

<u>Description</u>: Perceived Usefulness is a 6-item sub-scale measured at time point T2 (post-

intervention) to evaluate the usefulness of the intervention to help the participant to achieve their career-related goals using responses to items 6c, 9c through 9e, 10a, and 10b in the EVL Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4 points, and

5/Strongly Agree = 5 points.

Variable: PU\_T2\_1

<u>Label</u>: Perceived Usefulness Score at T2

Type: Numeric; Range = 1 to 5

Algorithm: PU\_T2\_1 = MEAN (EVL6c, EVL9c, EVL9d, EVL9e, EVL10a, EVL10b)

If all responses are missing, then PU\_T2\_1=Missing. Otherwise, consider mean of non-missing responses.

#### 1.1.4. ISSM Subscale 4: Overall Score

<u>Description</u>: The Overall Score is a 3-item sub-scale measured at time point T2 (post-intervention) to

evaluate the overall satisfaction with the workshops using responses to items 10c through 10e from the EVL Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4

points, and 5/Strongly Agree = 5 points.

<u>Variable</u>: OVERALL\_T2\_1

Label: Overall Score at T2

Type: Numeric; Range = 1 to 5

Algorithm: OVERALL T2 1 = MEAN (EVL10c, (6 - EVL10d), EVL10e)

If all responses are missing, then OVERALL \_T2\_1=Missing. Otherwise, consider mean of

non-missing responses.

## 1.1.5. Information Systems Success Model (ISSM) Score

Description: The ISSM Score is obtained by adding the four subscale scores defined above: IQ Score,

HQ Score, PU Score, and Overall Score.

Variable: ISSM\_T2\_1

<u>Label</u>: Information Systems Success Model Score at T2

Type: Numeric; Range = 1 to 5

 $\underline{Algorithm}: \quad ISSM\_T2\_1 = MEAN (IQ\_T2\_1, HQ\_T2\_1, PU\_T2\_1, OVERALL\_T2\_1).$ 

If all responses are missing, then ISSM\_T2\_1=Missing. Otherwise, consider mean of non-

missing responses.

#### 1.2. WORKSHOP COMPLETION

Workshop completion will be used in the assessment of intervention feasibility. The primary outcome for workshop completion will be measured using a binary outcome of Complete vs. Not Complete (1.2.2), but the number of completed workshops (1.2.1) is also defined to assess potential dose response of the workshop intervention on other outcomes.

#### 1.2.1. Number of Workshops Attended

<u>Description</u>: The participants' workshop attendance is recorded in items 3a, 3c, 4a, 4c, 5a, 5c, 6a, and

6c of the Workshop Tracking Information (WTI) form.

Variable: WSATTEND\_T2\_1

Label: Number of Workshops Attended at T2

Type: Numeric; Range = 0 to 4

Algorithm: WSATTEND\_T2\_1 = SUM (WTI3a, WTI3c, WTI4a, WTI4c, WTI5a, WTI5c, WTI6a, WTI6c)

If all responses are missing, then WSATTEND\_T2\_1=Missing. Otherwise, sum non-

missing responses. Note: WTI#c can only have a response if WTI#a=0.

## 1.2.2. Workshop Completion

<u>Description</u>: Workshop completion is defined as having attended at least two of the four workshop

sessions (50% completion).

Variable: WSCOMP\_T2\_1

<u>Label</u>: Workshop Completion at T2

<u>Type</u>: Numeric; Format: 0=Not Complete, 1=Complete, .=Missing

Algorithm: If WSATTEND T2 1 >= 2 then WSCOMP T2 1 = 1

Else if WSATTEND\_T2\_1 in (0, 1) then WSCOMP\_T2\_1=0

Else WSCOMP\_T2\_1 =  $\cdot$ 

#### 1.3. JOB SEEKING SELF-EFFICACY SCALE SCORE

Job seeking self-efficacy is defined as one's perceived ability and confidence to perform job search and application activities. Higher values indicate higher self-efficacy. This scale is measured at Baseline (T1) and the Month 8 Follow-up (T3).

## 1.3.1. Job Seeking Self-Efficacy Score at Baseline (T1)

<u>Description</u>: Job Seeking Self-Efficacy score at time point T1 (Baseline) is based on 12 items (52a

through 52f and 53a through 53f) from the BSL Questionnaire. Responses are scored on

the scale 1/Not at all confident = 1 point to 10/Very Confident = 10 points.

Variable: JOBSEEK T1 1

<u>Label</u>: Job-Seeking Self Efficacy Score at T1

Type: Numeric; Range = 1 to 10

Algorithm: JOBSEEK\_T1\_1 = MEAN(BSL52a, BSL52b, BSL52c, BSL52d, BSL52e, BSL52f, BSL53a,

BSL53b, BSL53c, BSL53d, BSL53e, BSL53f)

If all responses are missing, then JOBSEEK\_T1\_1=Missing. Otherwise, calculate the mean

of the non-missing responses.

#### 1.3.2. Job Seeking Self-Efficacy Score at Post-Intervention (T2)

Description: Job Seeking Self-Efficacy score at time point T2 (Post-Intervention) is based on 12 items

(13a through 13f and 14a through 14f) from the EVL Questionnaire. Responses are scored on the scale 1/Not at all confident = 1 point to 10/Very Confident = 10 points.

Variable: JOBSEEK\_T2\_1

Label: Job-Seeking Self Efficacy Score at T2

Type: Numeric; Range = 1 to 10

Algorithm: JOBSEEK\_T2\_1 = MEAN (EVL13a, EVL13b, EVL13c, EVL13d, EVL13e, EVL13f, EVL14a,

EVL14b, EVL14c, EVL14d, EVL14e, EVL14f)

If all responses are missing, then JOBSEEK\_T2\_1=Missing. Otherwise, calculate the mean

of the non-missing responses.

## 1.3.3. Job Seeking Self-Efficacy Score at Month 8 Follow-Up (T3)

Description: Job Seeking Self-Efficacy score at time point T3 (Month 8 follow-up) is based on 12 items

(52a through 52f and 53a through 53f) from the EXQ Questionnaire. Responses are scored on the scale 1/Not at all confident = 1 point to 10/Very Confident = 10 points.

Variable: JOBSEEK\_T3\_1

<u>Label</u>: Job-Seeking Self Efficacy Score at T3

Type: Numeric; Range = 1 to 10

Algorithm: JOBSEEK\_T3\_1 = MEAN (EXQ52a, EXQ52b, EXQ52c, EXQ52d, EXQ52e, EXQ52f, EXQ53a,

EXQ53b, EXQ53c, EXQ53d, EXQ53e, EXQ53f)

If all responses are missing, then JOBSEEK\_T3\_1=Missing. Otherwise, calculate the mean

of non-missing responses.

### 1.3.4. Change in Job Seeking Self-Efficacy Score from Baseline to Month 8 Follow-Up (T1T3)

<u>Description</u>: Difference between Job Seeking Self-Efficacy score at the Month 8 follow-up (T3) and

the score at Baseline (T1). If the Job Seeking Self-Efficacy score is missing at T3, then the

score from T2 is used to compute the change in score from T1.

Variable: JOBSEEK\_T1T3\_1

Label: Change in Job-Seeking Self Efficacy Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -9 to 9

Algorithm: If JOBSEEK\_T3\_1 not . then JOBSEEK\_T1T3\_1=JOBSEEK\_T3\_1 – JOBSEEK\_T1\_1

Else if JOBSEEK\_T3\_1=. then JOBSEEK\_T1T3\_1=JOBSEEK\_T2\_1 – JOBSEEK\_T1\_1

If JOBSEEK\_T1\_1 is missing, then JOBSEEK\_T1T3\_1=Missing. If JOBSEEK\_T2\_1 and

JOBSEEK T3 1 are missing, then JOBSEEK T1T3 1=Missing.

## 1.4. PROTEAN CAREER ATTITUDES SCALE (PCA) SCORE:

Protean career attitudes are defined as having self-direction in the pursuit of success in one's work. The scale (and the two sub scales) were measured at Baseline (T1) and the Month 8 follow-up (T3). Higher values indicate better attitudes.

#### 1.4.1. PCA Subscale 1: Self-Directed Attitudes Scale Score

## 1.4.1.1. Self-Directed Attitudes Score at Baseline (T1)

<u>Description</u>: Self-directed Attitudes Scale Score at time point T1 (Baseline) is based on four items

(75b, 75c, 75d, and 76a) from the BSL Questionnaire. Responses are scored as

1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3

points, 4/Agree = 4 points, and 5/Strongly Agree = 5 points.

Variable: SDA\_T1\_1

Label: Self-Directed Attitudes Scale Score at T1

Type: Numeric; Range = 1 to 5

Algorithm: SDA\_T1\_1 = MEAN (BSL75b, BSL75c, BSL 75d, BSL76a)

If all responses are missing, then SDA\_T1\_1=Missing. Otherwise, calculate the mean of

non-missing responses.

## 1.4.1.2. Self-Directed Attitudes Score at Month 8 Follow-Up (T3)

<u>Description</u>: Self-directed Attitudes Scale Score at time point T3 (Month 8 follow-up) is based on four

items (75b, 75c, 75d, and 76a) from the EXQ Questionnaire. Responses are recorded as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3

points, 4/Agree = 4 points, and 5/Strongly Agree = 5 points.

Variable: SDA T3 1

Label: Self-Directed Attitudes Scale Score at T3

Type: Numeric; Range = 1 to 5

<u>Algorithm</u>: SDA\_T3\_1 = MEAN (EXQ75b, EXQ75c, EXQ75d, EXQ76a)

If all responses are missing, then SDA\_T3\_1=Missing. Otherwise, calculate the mean of

non-missing responses.

## 1.4.1.3. Change in Self-Directed Attitudes Score from Baseline to Month 8 Follow-Up (T1T3)

Description: Difference between Self-Directed Attitudes score at time point T3 (Month 8 follow-up)

and time point T1 (Baseline)

Variable: SDA\_T1T3\_1

Label: Change in Self-Directed Attitudes Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -4 to 4

Algorithm:  $SDA_T1T3_1 = SDA_T3_1 - SDA_T1_1$ 

If SDA score at either time point is missing, then SDA T1T3 1=Missing.

#### 1.4.2. PCA Subscale 2: Values-Driven Attitudes Scale Score

## 1.4.2.1. Values-Driven Attitudes (VDA) Score at Baseline (T1)

Description: Values driven Attitudes Scale Score at time point T1 (Baseline) is based on 3 items (76b,

76c, and 76d) from the BSL Questionnaire. Response are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4

points, and 5/Strongly Agree = 5 points.

Variable: VDA\_T1\_1

<u>Label</u>: Values-Driven Attitudes Scale Score at T1

Type: Numeric; Range = 1 to 5

<u>Algorithm</u>:  $VDA_T1_1 = MEAN (BSL76b, BSL76c, BSL76d)$ 

If all responses are missing, then VDA\_T1\_1=Missing. Otherwise, calculate the mean of

non-missing responses.

### 1.4.2.2. Values-Driven Attitudes (VDA) Score at Month 8 Follow-Up (T3)

Description: Values driven Attitudes Scale Score at time point T3 (Month 8 follow-up) is based on 3

items (76b, 76c, and 76d) from the EXQ Questionnaire. Responses are scored as

1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3

points, 4/Agree = 4 points, and 5/Strongly Agree = 5 points

Variable: VDA T3 1

<u>Label</u>: Values-Driven Attitudes Scale Score at T3

Type: Numeric; Range = 1 to 5

<u>Algorithm</u>: VDA\_T3\_1 = MEAN (EXQ76b, EXQ76c, EXQ76d)

If all responses are missing, then VDA\_T3\_1=Missing. Otherwise, calculate the mean

ofnon-missing responses.

# 1.4.2.3. Change in Values-Driven Attitudes (VDA) Score from Baseline to Month 8 Follow-Up (T1T3)

<u>Description</u>: Difference between Values-Driven Attitudes Score at time point T3 (Month 8 follow-up)

from time point T1 (Baseline)

Variable: VDA\_T1T3\_1

<u>Label</u>: Change in Values Driven Attitudes Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -4 to 4

Algorithm:  $VDA_T1T3_1 = VDA_T3_1 - VDA_T1_1$ 

If VDA score at either time point is missing, then VDA\_T1T3\_1=Missing.

## 1.4.3. Scale: Protean Career Attitudes (PCA) Scale

### 1.4.3.1. Protean Career Attitudes (PCA) Score at Baseline (T1)

<u>Description</u>: The Protean Career Attitudes Score at T1 is obtained by adding the two subscale scores

defined above: SDA Score at T1 and VDA Score at T1.

Variable: PCA\_T1\_1

Label: Protean Career Attitudes Score at T1

Type: Numeric; Range = 1 to 5

Algorithm:  $PCA_T1_1 = MEAN (SDA_T1_1, VDA_T1_1)$ 

If either SDA or VDA score is missing, then PCA\_T1\_1=Missing.

## 1.4.3.2. Protean Career Attitudes (PCA) Score at Month 8 Follow-Up (T3)

<u>Description</u>: The Protean Career Attitudes Score at T3 is obtained by adding the two subscale scores

defined above: SDA Score at T3 and VDA Score at T3.

Variable: PCA\_T3\_1

Label: Protean Career Attitudes Score at T3

Type: Numeric; Range = 1 to 5

Algorithm: PCA\_T3\_1 = MEAN (SDA\_T3\_1, VDA\_T3\_1)

If either SDA or VDA score is missing, then PCA\_T3\_1=Missing.

# 1.4.3.3. Change in Protean Career Attitudes (PCA) Score from Baseline to Month 8 Follow-Up (T1T3)

<u>Description</u>: Difference between protean career attitudes score at time point T3 (Month 8 follow-up)

and time point T1 (Baseline)

Variable: PCA\_T1T3\_1

<u>Label</u>: Change in Protean Career Attitudes Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -4 to 4

Algorithm:  $PCA_T1T3_1 = PCA_T3_1 - PCA_T1_1$ .

If PCA score at either time point is missing, then PCA\_T1T3\_1=Missing.

## 2. SECONDARY OUTCOMES

#### 2.1. SELF-REPORTED EMPLOYMENT

The primary employment outcome is based on the change in the number of self-report hours worked per week from T1 to T3.

# 2.1.1. Change in Self-Reported Hours Worked Per Week from Baseline to Month 8 Follow-Up (T1T3)

<u>Description</u>: Change in hours worked per week from Baseline to Month 8 follow-up (T1 to T3)

Variable: EMPHOUR\_T1T3\_1

Label: Change in Hours Worked per Week from T1 to T3 (T3-T1)

Type: Numeric; Range = -99 to 99

Algorithm: If BSL9 = 0 then BSL27 = 0

If EXQ9 = 0 then EXQ27 = 0

 $EMPHOUR_T1T3_1 = EXQ27 - BSL27$ 

If hours work per week at either time point is missing, then EMPHOUR\_T1T3\_1=Missing.

## 2.2. SELF-REPORTED SEXUAL RISK BEHAVIORS

### 2.2.1. Self-Reported Sexual Risk Behavior at Baseline (T1)

Description: Sexual Risk behavior is measured using items 239 through 244 from the BSL

Questionnaire. Responses for each question are either Yes (1), No (0) or Missing (.). Risk

Behavior is defined as the mean of responses to the risk behavior questions.

Variable: RISK\_T1\_1

Label: Self-Reported Sexual Risk Behavior at T1

Type: Numeric; Range = 0 to 1

<u>Algorithm</u>: RISK\_T1\_1 = MEAN (BSL239, BSL240, BSL241, BSL242, BSL243, BSL244)

If responses for four or more individual risk behavior questions are missing, then RISK\_T1\_1 = Missing. Otherwise, calculate the mean of non-missing responses.

## 2.2.2. Self-Reported Sexual Risk Behavior at Baseline (T3)

<u>Description</u>: Sexual Risk behavior is measured using items 239 through 244 from the EXQ

Questionnaire. Responses for each question are either Yes (1), No (0) or Missing (.). Risk

Behavior is as the mean of responses to the risk behavior questions.

<u>Variable</u>: RISK\_T3\_1

Label: Self-Reported Sexual Risk Behavior at T3

Type: Numeric; Range = 0 to 1

Algorithm: RISK\_T3\_1 = MEAN (EXQ239, EXQ240, EXQ241, EXQ242, EXQ243, EXQ244)

If responses for four or more individual risk behavior questions are missing, then RISK\_T3\_1 = Missing. Otherwise, calculate the mean of non-missing responses.

## 2.2.3. Change in Self-Reported Risk Behavior from Baseline to Month 8 Follow-Up (T1T3)

<u>Description</u>: Change in Self-Reported Risk Behavior of a participant from Baseline to month 8 follow-

up (T1 to T3)

Variable: RISK\_T1T3\_1

<u>Label</u>: Change in Self-Reported Sexual Risk Behavior from T1 to T3 (T3-T1)

Type: Numeric; Range = -1 to 1

Algorithm:  $RISK_T1T3_1 = RISK_T3_1 - RISK_T1_1$ .

If risk behavior at either time point is missing, then RISK\_T1T3\_1 = Missing.

## 2.3. CHLAMYDIA INFECTIONS:

Chlamydia will be assessed at T1 (Baseline) and T3 (8-month follow-up) using urine, anal, and oral sample tests.

### 2.3.1. Chlamydia Result at Baseline (T1)

### 2.3.1.1. Chlamydia Result based on Oral Sample at T1

Description: The oral sample collection status is recorded in item 10a of the Biospecimen Collection

(BIC1) form and the oral swab Chlamydia result is recorded in item 1a of the

Biospecimen Results (BLR1) Form for Baseline (T1).

Variable: CH\_ORAL\_T1\_1

<u>Label</u>: Assessment of Chlamydia using an Oral Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC10a = 1 then CH ORAL T1 1 = [BLR1] BLR1a

Else if [BIC1] BIC10a=1 and [BLR1] BLR1a=. then CH\_ORAL\_T1\_1 = .U

Else if [BIC1] BIC10a=0 then CH\_ORAL\_T1\_1 = .N Else if [BIC1] BIC10a=9 then CH\_ORAL\_T1\_1 = .R Else if [BIC1] BIC10a=. then CH\_ORAL\_T1\_1 = .

## 2.3.1.2. Chlamydia Result based on Anal Sample at T1

<u>Description</u>: The anal sample collection status is recorded in item 11a of the BIC1 form and the anal

swab Chlamydia result is recorded in item 2a of the BLR1 Form for Baseline (T1).

Variable: CH\_ANAL\_T1\_1

<u>Label</u>: Assessment of Chlamydia using an Anal Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC11a = 1 then CH\_ANAL\_T1\_1 = [BLR1] BLR2a

Else if [BIC1] BIC11a=1 and [BLR1] BLR2a=. then CH\_ANAL\_T1\_1 = .U

Else if [BIC1] BIC11a=0 then ANAL\_CH\_T1\_1 = .N Else if [BIC1] BIC11a=9 then ANAL\_CH\_T1\_1 = .R Else if [BIC1] BIC11a=. then ANAL\_CH\_T1\_1 = .

### 2.3.1.3. Chlamydia Result based on Urine Sample at T1

Description: The urine sample collection status is recorded in item 12a of BIC1 form and the urine

Chlamydia result is recorded in item 3a of BLR1 Form for Baseline (T1).

Variable: CH\_URINE\_T1\_1

Label: Assessment of Chlamydia using a Urine Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

<u>Algorithm</u>: If [BIC1] BIC12a = 1 then CH\_URINE\_T1\_1 = [BLR1] BLR3a

Else if [BIC1] BIC12a=1 and [BLR1] BLR3a=. then CH\_URINE\_T1\_1 = .U

Else if [BIC1] BIC12a=0 then CH\_URINE\_T1\_1 = .N

Else if [BIC1] BIC12a=9 then CH\_URINE\_T1\_1 = .R Else if [BIC1] BIC12a=. then CH\_URINE\_T1\_1 = .

## 2.3.2. Chlamydia Result at Month 8 Follow-Up (T3)

#### 2.3.2.1. Chlamydia Result based on Oral Sample at T3

Description: The oral sample collection status is recorded in item 10a of the Biospecimen Collection

(BIC2) form and the oral swab Chlamydia result is recorded in item 1a of the

Biospecimen Results (BLR2) Form for 8-Month Follow-up (T3).

Variable: CH\_ORAL\_T3\_1

Label: Assessment of Chlamydia using an Oral Test T3

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC10a = 1 then CH\_ORAL\_T3\_1 = [BLR2] BLR1a

Else if [BIC2] BIC10a=1 and [BLR2] BLR1a=. then CH ORAL T3 1 = .U

Else if [BIC2] BIC10a=0 then CH\_ORAL\_T3\_1 = .N Else if [BIC2] BIC10a=9 then CH\_ORAL\_T3\_1 = .R Else if [BIC2] BIC10a=. then CH\_ORAL\_T3\_1 = .

#### 2.3.2.2. Chlamydia Result based on Anal Sample at T3

<u>Description</u>: The anal sample collection status is recorded in item 11a of the BIC2 form and the anal

swab Chlamydia result is recorded in item 2a of the BLR2 Form for the Month 8 follow-

up (T3).

Variable: CH\_ANAL\_T3\_1

Label: Assessment of Chlamydia using an Anal Test T3

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC11a = 1 then CH ANAL T3 1 = [BLR2] BLR2a

Else if [BIC2] BIC11a=1 and [BLR2] BLR2a=. then CH\_ANAL\_T3\_1 = .U

Else if [BIC2] BIC11a=0 then CH\_ANAL\_T3\_1 = .N Else if [BIC2] BIC11a=9 then CH\_ANAL\_T3\_1 = .R Else if [BIC2] BIC11a=. then CH\_ANAL\_T3\_1 = .

## 2.3.2.3. Chlamydia Result based on Urine Sample at T3

<u>Description</u>: The urine sample collection status is recorded in item 12a of BIC2 form and the urine

Chlamydia result is recorded in item 3a of BLR2 Form for Month 8 follow-up (T3).

Variable: CH\_URINE\_T3\_1

Label: Assessment of Chlamydia using a Urine Test T3

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC12a = 1 then CH\_URINE\_T3\_1 = [BLR2] BLR3a

Else if [BIC2] BIC12a=1 and [BLR2] BLR3a=. then CH\_URINE\_T3\_1 = .U

Else if [BIC2] BIC12a=0 then CH\_URINE\_T3\_1 = .N Else if [BIC2] BIC12a=9 then CH\_URINE\_T3\_1 = .R Else if [BIC2] BIC12a=. then CH\_URINE\_T3\_1 = .

## 2.3.3. Change in Chlamydia Result from Baseline to Month 8 Follow-Up (T1T3)

## 2.3.3.1. Change in Chlamydia Result based on Oral Samples at T1T3

Description: Change in Chlamydia oral sample result of a participant from Baseline to Month 8

follow-up (T1 to T3)

Variable: CH\_ORAL\_T1T3\_1

Label: Change in Chlamydia Oral Sample Result from T1 to T3 (T3-T1)

Type: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Anal Result,

-1=Positive to Negative

Algorithm: CH\_ORAL\_T1T3\_1 = CH\_ORAL\_T3\_1 - CH\_ORAL\_T1\_1

If measurement at either time point is missing, then CH\_ORAL\_T1T3\_1 = missing.

### 2.3.3.2. Change in Chlamydia Result based on Anal Samples at T1T3

Description: Change in Chlamydia anal sample result of a participant from Baseline to Month 8

follow-up (T1 to T3)

Variable: CH\_ANAL\_T1T3\_1

<u>Label</u>: Change in Chlamydia Anal Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Anal Result,

-1=Positive to Negative

<u>Algorithm:</u> CH\_ANAL\_T1T3\_1 = CH\_ANAL\_T3\_1 - CH\_ANAL\_T1\_1

If measurement at either time point is missing, then CH ANAL T1T3 1 = missing.

## 2.3.3.3. Change in Chlamydia Result based on Urine Samples at T1T3

Description: Change in Chlamydia urine sample result of a participant from Baseline to Month 8

follow-up (T1 to T3)

Variable: CH\_URINE\_T1T3\_1

<u>Label</u>: Change in Chlamydia Urine Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Anal Result,

-1=Positive to Negative

<u>Algorithm</u>: CH\_URINE\_T1T3\_1 = CH\_URINE\_T3\_1 - CH\_URINE\_T1\_1

If measurement at either time point is missing, then CH URINE T1T3 1 = missing.

#### 2.4. GONORRHEA INFECTIONS:

Gonorrhea will be assessed at T1 (Baseline) and T3 (8-Month follow-up) using urine, anal, and oral sample tests.

### 2.4.1. Gonorrhea Result at Baseline (T1)

#### 2.4.1.1. Gonorrhea Result based on Oral Sample at T1

<u>Description</u>: The oral sample collection status is recorded in item 10a of the BIC1 form and the oral

swab Gonorrhea result is recorded in item 1b of the BLR1 Form for Baseline (T1).

Variable: GN\_ORAL\_T1\_1

Label: Assessment of Gonorrhea using an Oral Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC10a = 1 then GN\_ORAL\_T1\_1 = [BLR1] BLR1b

Else if [BIC1] BIC10a=1 and [BLR1] BLR1b=. then GN ORAL T1 1 = .U

Else if [BIC1] BIC10a=0 then GN\_ORAL\_T1\_1 = .N Else if [BIC1] BIC10a=9 then GN\_ORAL\_T1\_1 = .R Else if [BIC1] BIC10a=. then GN\_ORAL\_T1\_1 = .

## 2.4.1.2. Gonorrhea Result based on Anal Sample at T1

<u>Description</u>: The anal sample collection status is recorded in item 11a of the BIC1 form and the anal

swab Gonorrhea result is recorded in item 2b of the BLR1 Form for Baseline (T1).

<u>Variable</u>: GN\_ANAL\_T1\_1

Label: Assessment of Gonorrhea using an Anal Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC11a = 1 then GN\_ANAL\_T1\_1 = [BLR1] BLR2b

Else if [BIC1] BIC11a=1 and [BLR1] BLR2b=. then GN\_ANAL\_T1\_1 = .U

Else if [BIC1] BIC11a=0 then GN\_ANAL\_T1\_1 = .N Else if [BIC1] BIC11a=9 then GN\_ANAL\_T1\_1 = .R Else if [BIC1] BIC11a=. then GN\_ANAL\_T1\_1 = .

## 2.4.1.3. Gonorrhea Result based on Urine Sample at T1

Description: The urine sample collection status is recorded in item 12a of BIC1 form and the urine

Gonorrhea result is recorded in item 3b of BLR1 Form for Baseline (T1).

<u>Variable</u>: GN\_URINE\_T1\_1

Label: Assessment of Gonorrhea using a Urine Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC12a = 1 then GN URINE T1 1 = [BLR1] BLR3b

Else if [BIC1] BIC12a=1 and [BLR1] BLR3b=. then GN URINE T1 1 = .U

Else if [BIC1] BIC12a=0 then GN\_URINE\_T1\_1 = .N Else if [BIC1] BIC12a=9 then GN\_URINE\_T1\_1 = .R Else if [BIC1] BIC12a=. then GN\_URINE\_T1\_1 = .

### 2.4.2. Gonorrhea Result at Month 8 Follow-Up (T3)

### 2.4.2.1. Gonorrhea Result based on Oral Sample at T3

<u>Description</u>: The oral sample collection status is recorded in item 10a of the BIC2 form and the oral

swab Gonorrhea result is recorded in item 1b of the BLR2 Form for 8-Month follow-up

(T3).

Variable: GN\_ORAL\_T3\_1

Label: Assessment of Gonorrhea using an Oral Test T3

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC10a = 1 then GN\_ORAL\_T3\_1 = [BLR2] BLR1b

Else if [BIC2] BIC10a=1 and [BLR2] BLR1b=. then GN ORAL T3 1 = .U

Else if [BIC2] BIC10a=0 then GN\_ORAL\_T3\_1 = .N Else if [BIC2] BIC10a=9 then GN\_ORAL\_T3\_1 = .R Else if [BIC2] BIC10a=. then GN\_ORAL\_T3\_1 = .

## 2.4.2.2. Gonorrhea Result based on Anal Sample at T3

<u>Description</u>: The anal sample collection status is recorded in item 11a of the BIC2 form and the anal

swab Gonorrhea result is recorded in item 2b of the BLR2 Form for the Month 8 follow-

up (T3).

Variable: GN ANAL T3 1

Label: Assessment of Gonorrhea using an Anal Test T3

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC11a = 1 then GN\_ANAL\_T3\_1 = [BLR2] BLR2b

Else if [BIC2] BIC11a=1 and [BLR2] BLR2b=. then GN\_ANAL\_T3\_1 = .U

Else if [BIC2] BIC11a=0 then GN\_ANAL\_T3\_1 = .N Else if [BIC2] BIC11a=9 then GN\_ANAL\_T3\_1 = .R Else if [BIC2] BIC11a=. then GN\_ANAL\_T3\_1 = .

#### 2.4.2.3. Gonorrhea Result based on Urine Sample at T3

<u>Description</u>: The urine sample collection status is recorded in item 12a of BIC2 form and the urine

Gonorrhea result is recorded in item 3b of BLR2 Form for Month 8 follow-up (T3).

Variable: GN\_URINE\_T3\_1

<u>Label</u>: Assessment of Gonorrhea using a Urine Test T3

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC12a = 1 then GN\_URINE\_T3\_1 = [BLR2] BLR3b

Else if [BIC2] BIC12a=1 and [BLR2] BLR3b=. then GN\_URINE\_T3\_1 = .U

Else if [BIC2] BIC12a=0 then GN\_URINE\_T3\_1 = .N Else if [BIC2] BIC12a=9 then GN\_URINE\_T3\_1 = .R

Else if [BIC2] BIC12a=. then GN\_URINE\_T3\_1 = .

## 2.4.3. Change in Gonorrhea Result from Baseline to Month 8 Follow-Up (T1T3)

## 2.4.3.1. Change in Gonorrhea Result based on Oral Samples at T1T3

<u>Description</u>: Change in Gonorrhea oral sample result of a participant from Baseline to Month 8

follow-up (T1 to T3)

Variable: GN\_ORAL\_T1T3\_1

<u>Label</u>: Change in Gonorrhea Oral Sample Result from T1 to T3 (T3-T1)

Type: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Oral Result, -

1=Positive to Negative

Algorithm: GN\_ORAL\_T1T3\_1 = GN\_ORAL\_T3\_1 - GN\_ORAL\_T1\_1

If measurement at either time point is missing, then GN ORAL T1T3 1 = missing.

## 2.4.3.2. Change in Gonorrhea Result based on Anal Samples at T1T3

Description: Change in Gonorrhea anal sample result of a participant from Baseline to Month 8

follow-up (T1 to T3)

Variable: GN\_ANAL\_T1T3\_1

<u>Label</u>: Change in Gonorrhea Anal Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Anal Result, -

1=Positive to Negative

Algorithm: GN\_ANAL\_T1T3\_1 = GN\_ANAL\_T3\_1 - GN\_ANAL\_T1\_1

If measurement at either time point is missing, then GN ANAL T1T3 1 = missing.

## 2.4.3.3. Change in Gonorrhea Result based on Urine Samples at T1T3

Description: Change in Gonorrhea urine sample result of a participant from Baseline to Month 8

follow-up (T1 to T3)

Variable: GN\_URINE\_T1T3\_1

Label: Change in Gonorrhea Urine Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea urine result, -

1=Positive to Negative

Algorithm: GN\_URINE\_T1T3\_1 = GN\_URINE\_T3\_1 - GN\_URINE\_T1\_1

If measurement at either time point is missing, then GN\_URINE\_T1T3\_1 = missing.

### 2.5. REACTIVE HIV TEST

<u>Description</u>: Testing for HIV is conducted at Baseline (T1) and Month 8 follow-up (T3) and indicates

whether or not the test result was reactive or non-reactive. The reactive HIV testing

result for T3 is recorded in item 1a of the BIC2 form.

Variable: HIVREAC\_T3\_1

Label: Reactive HIV Test Result at T3.

<u>Type</u>: Numeric; Format: 0=Non-Reactive, 1=Reactive, .U=Unknown, .N=Not Collected,

.R=Refused, .=Missing

Algorithm: If [BIC2] BIC1=1 then HIVREAC\_T3\_1= [BIC2] BIC1a

Else if [BIC2] BIC1=1 and [BIC2] BIC1a=. then HIVREAC\_T3\_1=.U

Else if [BIC2] BIC1=0 then HIVREAC T3 1 1 = .N

Else if [BIC2] BIC1=9 and [BIC2] BIC1a=9 then HIVREAC\_T3\_1=.R Else if [BIC2] BIC1=. and [BIC2] BIC1a=. then HIVREAC\_T3\_1=.

# Statistical Analysis Plan: Work2Prevent – Phase 3

**PROTOCOL:** ATN 151: Work2Prevent: Employment as HIV prevention

for young men who have sex with men (YMSM) and young

transgender women (YTW)

PROTOCOL DATE: May 23, 2017

Revised August 5, 2019

PROTOCOL VERSION: 5.1

CLINICALTRIALS.GOV ID: NCT03313310

**SPONSOR:** The Eunice Kennedy Shriver National Institute of Child

Health and Human Development (NICHD)

with co-funding from:

National Institute on Drug Abuse (NIDA),

National Institute of Mental Health (NIMH), and National Institute on Minority Health and Health

Disparities (NIMHD)

SAP DATE: December 13, 2019

SAP VERSION: 2.0

SAP PREPARED BY: ATN Coordinating Center

**Collaborative Studies Coordinating Center** 

**Department of Biostatistics** 

The University of North Carolina at Chapel Hill 123 W. Franklin Street, Suite 450, CB# 8030

Chapel Hill, NC 27599-8030

AUTHORS: Myra A. Carpenter, PhD

Micah McCumber, MS Cara M. Nordberg, MPH Justin Demonte, BS Betty Rupp, MPH

# SIGNATURE PAGE

| Name | Role | Signature | Date |
|----------------|------------------------|-----------|------|
| Lisa Strader | ATN CC Co-Investigator | | |
| Brandon Hill | Principal Investigator | | |
| Darnell Motley | Site Investigator | | |

# **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 7 |
|----|-------------------------------------------------------------------|-----|
| | 1.1. OBJECTIVES AND RESEARCH HYPOTHESES | 7 |
| 2. | STUDY METHODS | 7 |
| | 2.1. Study Design | 7 |
| | 2.2. Study Population | 7 |
| | 2.3. Sample Size Information | 8 |
| 3. | ANALYSIS POPULATIONS | 8 |
| | 3.1. PER PROTOCOL POPULATION ERROR! BOOKMARK NOT DEFIN | ED. |
| 4. | STUDY ASSESSMENTS | 9 |
| | 4.1. Primary Outcomes | 9 |
| | 4.1.1. Information Systems Success Model Score (T2) | 9 |
| | 4.1.2. Workshop Completion (T2) | 9 |
| | 4.1.3. Change in Job-Seeking Self-Efficacy Scale Score (T1 to T3) | 9 |
| | 4.1.4. Change in Protean Career Attitudes Scale Score (T1 to T3) | 10 |
| | 4.2. Secondary Outcomes | 10 |
| | 4.2.1. Change in Self-Reported Hours Worked Per Week (T1 to T3) | 10 |
| | 4.2.2. Change in Self-Reported Sexual Risk Behaviors (T1 to T3) | 10 |
| | 4.2.3. Change in Chlamydia Test Result (T1 to T3) | 11 |
| | 4.2.4. Change in Gonorrhea Test Result (T1 to T3) | 11 |
| | 4.2.5. Reactive HIV Test (T3) | 11 |
| 5. | STATISTICAL ANALYSIS | 11 |
| | 5.1. GENERAL CONSIDERATIONS | 11 |
| | 5.2. Missing Data | 11 |
| | 5.3. Subject Disposition Analyses | 12 |
| | 5.4. Analysis of Primary Outcomes | 12 |
| | 5.5. Analysis of Secondary Outcomes | 12 |
| | 5.6. ANALYSIS OF SAFETY EVENTS | 12 |
| RE | FERENCES | 13 |
| ΑP | PENDIX | 14 |
| 1. | PRIMARY OUTCOMES | 14 |
| | 1.1. INFORMATION SYSTEMS SUCCESS MODEL (ISSM) SCALE | 14 |
|---|---|---|
| | 1.1.1. ISSM Subscale 1: Information Quality (IQ) Score | 14 |
| | 1.1.2. ISSM Subscale 2: Handbook Quality (HQ) Score | 14 |
| | 1.1.3. ISSM Subscale 3: Perceived Usefulness (PU) Score | 15 |
| | 1.1.4. ISSM Subscale 4: Overall Score | 15 |
| | 1.1.5. Information Systems Success Model (ISSM) Score | 16 |
| | 1.2. WORKSHOP COMPLETION | 16 |
| | 1.2.1. Number of Workshops Attended | 16 |
| | 1.2.2. Workshop Completion | 16 |
| | 1.3. JOB SEEKING SELF-EFFICACY SCALE SCORE | 17 |
| | 1.3.1. Job Seeking Self-Efficacy Score at Baseline (T1) | 17 |
| | 1.3.2. Job Seeking Self-Efficacy Score at Post-Intervention (T2) | 17 |
| | 1.3.3. Job Seeking Self-Efficacy Score at Month 3 Follow-Up (T3) | 18 |
| | 1.3.4. Change in Job Seeking Self-Efficacy Score from Baseline to Month 3 Follow (T1T3) | - |
| | 1.4. PROTEAN CAREER ATTITUDES SCALE (PCA) SCORE: | 19 |
| | 1.4.1. PCA Subscale 1: Self-Directed Attitudes (SDA) Scale Score | 19 |
| | 1.4.2. PCA Subscale 2: Values-Driven Attitudes Scale Score | 20 |
| | 1.4.3. Scale: Protean Career Attitudes (PCA) Scale | 21 |
| 2. | SECONDARY OUTCOMES | 23 |
| | 2.1. SELF-REPORTED EMPLOYMENT | 23 |
| | 2.1.1. Change in Self-Reported Hours Worked Per Week from Baseline to Month Follow-Up (T1T3) | |
| | 2.2. SELF-REPORTED SEXUAL RISK BEHAVIORS | 23 |
| | 2.2.1. Self-Reported Sexual Risk Behavior at Baseline (T1) | 23 |
| | 2.2.2. Self-Reported Sexual Risk Behavior at Baseline (T3) | 24 |
| | 2.2.3. Change in Self-Reported Risk Behavior from Baseline to Month 3 Follow-U (T1T3) | |
| | 2.3. CHLAMYDIA INFECTIONS: | |
| | 2.3.1. Chlamydia Result at Baseline (T1) | 24 |
| | 2.3.2. Chlamydia Result at Month 3 Follow-Up (T3) | |
| | 2.3.3. Change in Chlamydia Result from Baseline to Month 3 Follow-Up (T1T3) | 27 |

| 2.4. GONORRHEA INFECTIONS: | 28 |
|---|---|
| 2.4.1. Gonorrhea Result at Baseline (T1) | 28 |
| 2.4.2. Gonorrhea Result at Month 3 Follow-Up (T3) | 29 |
| 2.4.3. Change in Gonorrhea Result from Baseline to Month 3 Follow-Up (T1T3) | 31 |
| 2.5. REACTIVE HIV TEST | 32 |

#### LIST OF ABBREVIATIONS

AIDS Acquired Immunodeficiency Syndrome

ATN Adolescent Medicine Trials Network for HIV/AIDS Interventions

CAI Condomless Anal Intercourse CC ATN Coordinating Center

CSCC Collaborative Studies Coordinating Center

HIV Human Immunodeficiency Virus

HQ Handbook Quality IQ Information Quality

ISSM Information Systems Success Model

JSS Job-Seeking Self-Efficacy
MSM Men who have Sex with Men

NICHD Eunice Kennedy Shriver National Institute of Child Health and Human Development

NIDA National Institute on Drug Abuse
NIMH National Institute of Mental Health

NIMHD National Institute on Minority Health and Health Disparities

PCA Protean Career Attitudes
PU Perceived Usefulness
SDA Self-Directed Attitudes

STI Sexually Transmitted Infection

T1 Baseline Visit

T2 Post-Intervention Visit at 0-2 weeks post-intervention
T3 Follow-up Visit at 3-months (±2 weeks) post-intervention

VDA Values-Driven Attitudes

W2P Work2Prevent

YMSM Young Men who have Sex with Men

YTW Young Transgender Women

#### 1. INTRODUCTION

Work2Prevent (W2P) is a study designed to adapt, tailor, and pilot-test a novel social and structural-level HIV intervention for Young Men who have Sex with Men (YMSM) and Young Transgender Women (YTW) of color aimed at increasing economic stability (i.e., employment) through youth empowerment, increased self-efficacy, and decreased HIV risk behaviors (i.e., sex work) associated with social and economic marginalization. This document provides details of the planned statistical analysis for Phase 3 of intervention.

# 1.1. Objectives and Research Hypotheses

The primary objective of Phase 3 is to pilot-test a intervention among up to 40 at-risk YMSM and YTW of color to evaluate feasibility and acceptability. Investigators hypothesize the intervention will increase job self-efficacy and readiness, as well as decrease HIV risk behaviors and STI and HIV infections.

#### 2. STUDY METHODS

## 2.1. Study Design

W2P is a single-arm longitudinal pre and post study of a social and structural-level employment intervention to evaluate feasibility, acceptability, and satisfaction of the intervention program, and preliminary efficacy for study outcomes assessed at Baseline (T1), Post-Intervention (T2, 0 to 2 weeks post workshop completion), and 3-Month Follow-up (±2 weeks) (T3). The study employment intervention is comprised of four structured workshops presented over a 2-day period.

The study aims to enroll up to 40 at-risk YMSM and YTW of color over a 6-month period. The intervention workshops will be completed within 4 weeks of enrollment. Each participant will then be assessed 3-months (±2 weeks) post-intervention.

Study outcomes include: (1) job self-efficacy and readiness; (2) HIV risk behaviors; (3) employment; and (4) STI and HIV infections.

## 2.2. Study Population

All intervention study participants are Black, African American, Hispanic, or Latinx males, including transgender women (those assigned male at birth), ages 16-24, who identify as either an (1) MSM or gay or bisexual man or as a (2) transgender woman or transsexual male-to-female or transwoman.

## Participant Inclusion Criteria:

- 1. Being male or assigned male at birth (YTW)
- 2. Identifying as YMSM, gay bisexual man, transgender woman, or transwoman
- 3. Identifying as African American, Black, Hispanic, or Latinx
- 4. 16-24 years old
- 5. English-speaking (primary)
- 6. Currently unemployed but seeking employment, or employed only part-time (average of 35 hours or less per week)
- 7. Able to attend a 4-session employment program over 2 days
- 8. Did not participate in Phase 2 pilot

## Participant Exclusion Criteria:

- 1. Individuals identifying as non-Hispanic White
- 2. Individuals not assigned male at birth

# 2.3. Sample Size Information

This study aims to enroll up to 40 participants. Given the exploratory nature of this study and limited access to this population, a power calculation was not performed. A repeated measures design was chosen to reduce the variability in the estimate of the treatment effect, at the expense of having a comparison group. In addition, practice or fatigue effects from repetition may affect certain outcomes (e.g. protean career attitudes scale and subscales). This trade-off was appropriate given the exploratory nature of a pilot study and the limited access to the study population.

#### 3. ANALYSIS POPULATIONS

Only participants who are enrolled at Baseline (complete the T1 survey) will be included in the primary and secondary analyses. Screen-failures will not be included in these analyses.

## 3.1. Intent-to-Treat Population

All participants who completed T3 will be included in intent-to-treat analyses involving variables measuring changes from T1 to T3 (see sections 4.1.3-4.1.4 and 4.2.1-4.2.5 below). All participants who completed at least one workshop will be included in intent-to-treat analyses involving workshop evaluation and workshop completion variables (see sections 4.1.1, 4.1.2 below). This population will form the basis for both the primary and secondary analyses of the efficacy and safety endpoints.

## 3.2. Per Protocol Population

Youth who attend at least two of the four planned intervention workshops and complete T3 will comprise the per protocol population. This population will form the basis for both the primary and secondary analyses of the efficacy and safety endpoints.

#### 4. STUDY ASSESSMENTS

| Study Assessments | Pre-Screening | Baseline<br>(T1) | Post-<br>Intervention (T2) | 3-Month<br>Follow-Up (T3) |
|---|---|---|---|---|
| Screener Survey (SCR) | X | | | |
| Eligibility Form (ELG) | | Χ | | |
| Baseline Survey (BSL) | | Χ | | |
| Biospecimen Collection Form (BIC) | | Х | | Х |
| Biospecimen Lab Results<br>Form (BLR) | | Х | | Х |
| Workshop Tracking (WTI) | | | X | |
| Workshop Evaluation (EVL) | | | X | |
| Exit Visit Survey (EXQ) | | | | X |

# 4.1. Primary Outcomes

## 4.1.1. Information Systems Success Model Score (T2)

The Information Systems Success Model (ISSM) will be used to assess for intervention acceptability and satisfaction. The 21-item scale measures four sub-domains: information quality, handbook quality, perceived usefulness, and overall satisfaction. Every item is scored on a 1 to 5 scale, with 1 being "Strongly Disagree" and 5 being "Strongly Agree". Responses are averaged within each sub-domain to produce four sub-domain scores. The four sub-domain scores are then averaged to produce an overall ISSM score (range: 1 to 5; higher scores indicate higher acceptability/satisfaction). This scale has been adapted from Horvath et al.<sup>1</sup>

# 4.1.2. Workshop Completion (T2)

Workshop completion will be used to assess for intervention feasibility. The outcome of intervention completion is defined as having attended at least two of the four workshop sessions and is measured by tracking participant attendance. Workshop completion may also be defined as the number of workshop sessions attended for use in exploratory analyses.

## 4.1.3. Change in Job-Seeking Self-Efficacy Scale Score (T1 to T3)

Job seeking self-efficacy is defined as one's perceived ability and confidence to perform job search and application activities. The 12-item Job Seeking Self-Efficacy (JSS) scale by Barlow, Wright, & Cullen<sup>2</sup> uses response values on a 1 to 10 score, with 1 being "Not At All Confident"

and 10 being "Very Confident". Reponses are averaged to yield a total score, with higher scores indicating higher self-efficacy. Change in JSS will be calculated by subtracting the JSS score at baseline (T1) from the JSS score at the 3-month follow-up (T3) (range: -9 to +9; negative change indicates decreased self-efficacy, while positive change indicates increased self-efficacy).

# 4.1.4. Change in Protean Career Attitudes Scale Score (T1 to T3)

Protean career attitudes (PCAs) are defined as having self-direction in the pursuit of success in one's work. PCAs have previously been found to be associated with positive career satisfaction and self-perceived success.<sup>3</sup> The validated 7-item scale by Porter, Woo, & Tak<sup>4</sup> measures two sub-domains: self-directed attitudes and value-driven attitudes. Every item is scored on a 1 to 5 scale, with 1 being "Strongly Disagree" and 5 being "Strongly Agree". Responses are averaged within each sub-domain to produce two sub-domain scores, which are then averaged to produce an overall PCA score. Change in PCA score will be calculated by subtracting the score at baseline (T1) from the score at the 3-month follow-up (T3) (range: -4 to +4; negative change indicates decreased PCAs, while positive change indicates increased PCAs).

# 4.2. Secondary Outcomes

# 4.2.1. Change in Self-Reported Hours Worked Per Week (T1 to T3)

Hours worked per week will be self-reported at baseline and at the 3-month follow-up visit as any value between 0 and 99. Change in hours worked per week will be calculated by subtracting the baseline (T1) value from the 3-month follow-up (T3) value. Negative change indicates fewer hours worked per week, while positive change indicates more hours worked per week.

# 4.2.2. Change in Self-Reported Sexual Risk Behaviors (T1 to T3)

Sexual risk behaviors will be measured using six yes or no (1 or 0) items assessing for engagement in the following behaviors during the 3 months prior to baseline (T1) and 3-month follow-up (T3) assessments:

- 1. Condomless anal intercourse (CAI) with male partner of unknown HIV status
- 2. Anal intercourse with ≥3 males
- 3. Sex with male partner with a Sexually Transmitted Infection (STI)
- 4. CAI with HIV+ male partner
- 5. Anal intercourse with condom failure
- 6. Transactional sex work involvement

Responses will be averaged at each assessment. Change in sexual risk behaviors will be calculated by subtracting the average at baseline from the average at the 3-month follow-up (range: -1 to +1; negative change indicates fewer sexual risk behaviors, while positive change indicates more sexual risk behaviors).

# 4.2.3. Change in Chlamydia Test Result (T1 to T3)

Chlamydia infections will be assessed at baseline and 3-month follow up using oral, anal, and urine samples. Each of the three tests yields a positive (1) or negative (0) result. Change in test result will be calculated by subtracting the baseline result from the 3-month follow-up result. Oral, anal, and urine tests will be treated as separate outcomes.

# 4.2.4. Change in Gonorrhea Test Result (T1 to T3)

Gonorrhea infections will be assessed at baseline and 3-month follow up using oral, anal, and urine samples. Each of the three tests yields a positive (1) or negative (0) result. Change in test result will be calculated by subtracting the baseline result from the 3-month follow-up result. Oral, anal, and urine tests will be treated as separate outcomes.

## 4.2.5. Reactive HIV Test (T3)

Testing for HIV will be assessed at baseline and 3-month follow up. The test yields a reactive (1) or non-reactive (0) result. The outcome for reactive HIV test will use the T3 test result.

#### 5. STATISTICAL ANALYSIS

#### 5.1. General Considerations

The analytic plan is designed to determine preliminary efficacy of the intervention by comparing pre and post assessments of employment and sexual risk behaviors. Descriptive statistics will be used to analyze the proportions and central tendencies for participant sociodemographic covariates collected in the surveys. We will first generate frequencies, means, and other measures of central tendency as appropriate to describe our sample and outcomes at each of the three time points (baseline, post-intervention, and 3-month follow-up).

Changes in primary and secondary outcomes between baseline and 3-month follow-up will be assessed using paired t-tests for continuous variables and McNemar's test for matched categorical variables. We will use standard diagnostic tools to assess the appropriateness of the normality assumption (e.g., QQ-plots) and, if approximate normality of the residuals is not tenable, a non-parametric test for continuous paired data, i.e., Wilcoxon sign rank test will be used. All hypothesis testing will be done at an alpha-level of 0.1, given the exploratory nature of the study.

#### 5.2. Missing Data

Missing responses to survey questions will be excluded and non-missing data will be used to compute the primary and secondary outcomes. If all components for an outcome are missing, then the outcome will be considered missing. For those outcomes with unique missing data rules, the handling of missing data for each individual outcome are described in the appendix.

Missing data patterns will be explored prior to the analysis of the primary and secondary outcomes.

# **5.3. Subject Disposition Analyses**

Number of participants pre-screened, screened, eligible, discontinued, and included in the per protocol analysis population will be reported. In addition, the number of participants completing each visit (T1, T2 and T3) and the reasons for patient discontinuation will be tabulated.

# 5.4. Analysis of Primary Outcomes

Primary outcomes for analyses include Information Systems Success Model score, workshop completion, change in Job-Seeking Self Efficacy Scale score, Protean Career Attitudes Scale score, change in Self-Directed Attitudes Scale score, and change in Values-Driven Attitudes Scale score. Details about these outcomes are described in Section 4.1.

Univariate analyses will be performed as described in Section 5.1. To the extent that data allows, multivariable analyses will adjust for sociodemographic characteristics, workshop attendance, baseline employment status, and study completeness. Analytical models will include linear regression or generalized linear models for continuous outcomes and logistic regression for binary and categorical outcomes.

#### **5.5. Analysis of Secondary Outcomes**

Secondary outcomes for analyses include change in self-reported hours worked per week, change in self-reported sexual risk behavior, change in chlamydia test results, change in gonorrhea test results, and reactive HIV test result. Details about these outcomes are described in Section 4.2.

Univariate analyses will be performed as described in Section 5.1. Multivariable analyses will adjust for sociodemographic characteristics, workshop attendance, baseline employment status, and study completeness. Analytical models will include linear regression or generalized linear models for continuous outcomes and logistic regression for binary and categorical outcomes.

# 5.6. Analysis of Safety Events

Safety events will be recorded for participants as needed throughout the study. The number of participants experiencing each safety event will be summarized by severity grade, relationship to study, and action taken. All safety events will be provided in the safety events data listing. Withdrawals due to safety events will also be reported.

#### **REFERENCES**

- 1. Horvath KJ, Oakes MJ, Rosser SBR, Danilenko G, Vezina H, Amico RK, Williams ML, Simoni J. Feasibility, Acceptability and Preliminary Efficacy of an Online Peer-to-Peer Social Support ART Adherence Intervention. AIDS Behav., 2013; 17:2031-2044.
- 2. Barlow J, Wright C, Cullen L. *A job-seeking self-efficacy scale for people with physical disabilities: preliminary development and psychometric testing.* Br J Guid Counc., 2002; 30:1, 37-53.
- 3. Volmer J, Spurk D. *Protean and boundaryless career attitudes: relationships with subjective and objective career success.* J Labor Mark Res., 2011; 43:207-218.
- 4. Porter C, Woo SE, Tak J. *Developing and Validating Short Form Protean and Boundaryless Career Attitudes Scales*. J Career Assess., 2016; 24(1):162-181.

## 1. PRIMARY OUTCOMES

# 1.1. INFORMATION SYSTEMS SUCCESS MODEL (ISSM) SCALE

The Information Systems Success Model (ISSM) scale has been adapted from Horvath et al.<sup>1</sup> to assess intervention acceptability and satisfaction. The scale evaluates four sub-domains: information quality, system quality, perceived usefulness, and overall satisfaction. For each of the calculated scores, higher values indicate better participant-assessed quality.

# 1.1.1. ISSM Subscale 1: Information Quality (IQ) Score

<u>Description</u>: Information Quality is a 6-item sub-scale measured at time point T2 (post-intervention)

to evaluate ease of comprehension, credibility, clarity, and accuracy of the information provided through the intervention using responses to items 7a through 7e and 8a in the Evaluation (EVL) Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4 points, and

5/Strongly Agree = 5 points.

Variable: IQ\_T2\_1

<u>Label:</u> Information Quality Score at T2

Type: Numeric; Range = 1 to 5

<u>Algorithm:</u> IQ\_T2\_1 = MEAN (EVL7a, EVL7b, EVL7c, EVL7d, EVL7e, EVL8a)

If all responses are missing, then then IQ\_T2\_1=Missing. Otherwise, consider mean of

non-missing responses.

## 1.1.2. ISSM Subscale 2: Handbook Quality (HQ) Score

<u>Description</u>: Handbook Quality is a 6-item sub-scale measured at time point T2 (post-intervention) to

evaluate user friendliness and appeal of the workshop handbook provided through the

intervention using responses to items 8b through 8e, 9a, and 9b in the EVL

Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4 points, and 5/Strongly

Agree = 5 points.

<u>Variable</u>: HQ\_T2\_1

Label: Handbook Quality Score at T2

Type: Numeric; Range = 1 to 5

Algorithm: HQ\_T2\_1 = MEAN (EVL8b, EVL8c, EVL8d, EVL8e, EVL9a, EVL9b)

If all responses are missing, then HQ\_T2\_1=Missing. Otherwise, consider mean of non-missing responses.

# 1.1.3. ISSM Subscale 3: Perceived Usefulness (PU) Score

<u>Description</u>: Perceived Usefulness is a 6-item sub-scale measured at time point T2 (post-

intervention) to evaluate the usefulness of the intervention to help the participant to achieve their career-related goals using responses to items 6c, 9c through 9e, 10a, and 10b in the EVL Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4 points, and

5/Strongly Agree = 5 points.

Variable: PU\_T2\_1

<u>Label</u>: Perceived Usefulness Score at T2

Type: Numeric; Range = 1 to 5

Algorithm: PU\_T2\_1 = MEAN (EVL6c, EVL9c, EVL9d, EVL9e, EVL10a, EVL10b)

If all responses are missing, then PU\_T2\_1=Missing. Otherwise, consider mean of non-missing responses.

#### 1.1.4. ISSM Subscale 4: Overall Score

<u>Description</u>: The Overall Score is a 3-item sub-scale measured at time point T2 (post-intervention) to

evaluate the overall satisfaction with the workshops using responses to items 10c through 10e from the EVL Questionnaire. Responses are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4

points, and 5/Strongly Agree = 5 points.

<u>Variable</u>: OVERALL\_T2\_1

Label: Overall Score at T2

Type: Numeric; Range = 1 to 5

Algorithm: OVERALL T2 1 = MEAN (EVL10c, (6 - EVL10d), EVL10e)

If all responses are missing, then OVERALL \_T2\_1=Missing. Otherwise, consider mean of

non-missing responses.

# 1.1.5. Information Systems Success Model (ISSM) Score

Description: The ISSM Score is obtained by adding the four subscale scores defined above: IQ Score,

HQ Score, PU Score, and Overall Score.

Variable: ISSM\_T2\_1

<u>Label</u>: Information Systems Success Model Score at T2

Type: Numeric; Range = 1 to 5

 $\underline{Algorithm}: \quad ISSM\_T2\_1 = MEAN (IQ\_T2\_1, HQ\_T2\_1, PU\_T2\_1, OVERALL\_T2\_1).$ 

If all responses are missing, then ISSM\_T2\_1=Missing. Otherwise, consider mean of non-

missing responses.

#### 1.2. WORKSHOP COMPLETION

Workshop completion will be used in the assessment of intervention feasibility. The primary outcome for workshop completion will be measured using a binary outcome of Complete vs. Not Complete (1.2.2), but the number of completed workshops (1.2.1) is also defined to assess potential dose response of the workshop intervention on other outcomes.

#### 1.2.1. Number of Workshops Attended

<u>Description</u>: The participants' workshop attendance is recorded in items 3a, 3c, 4a, 4c, 5a, 5c, 6a, and

6c of the Workshop Tracking Information (WTI) form.

Variable: WSATTEND\_T2\_1

Label: Number of Workshops Attended at T2

Type: Numeric; Range = 0 to 4

Algorithm: WSATTEND\_T2\_1 = SUM (WTI3a, WTI3c, WTI4a, WTI4c, WTI5a, WTI5c, WTI6a, WTI6c)

If all responses are missing, then WSATTEND\_T2\_1=Missing. Otherwise, sum non-

missing responses. Note: WTI#c can only have a response if WTI#a=0.

# 1.2.2. Workshop Completion

<u>Description</u>: Workshop completion is defined as having attended at least two of the four workshop

sessions (50% completion).

Variable: WSCOMP\_T2\_1

<u>Label</u>: Workshop Completion at T2

<u>Type</u>: Numeric; Format: 0=Not Complete, 1=Complete, .=Missing

Algorithm: If WSATTEND T2 1 >= 2 then WSCOMP T2 1 = 1

Else if WSATTEND\_T2\_1 in (0, 1) then WSCOMP\_T2\_1=0

Else WSCOMP\_T2\_1 = .

#### 1.3. JOB SEEKING SELF-EFFICACY SCALE SCORE

Job seeking self-efficacy is defined as one's perceived ability and confidence to perform job search and application activities. Higher values indicate higher self-efficacy. This scale is measured at Baseline (T1) and the Month 3 Follow-up (T3).

# 1.3.1. Job Seeking Self-Efficacy Score at Baseline (T1)

<u>Description</u>: Job Seeking Self-Efficacy score at time point T1 (Baseline) is based on 12 items (52a

through 52f and 53a through 53f) from the BSL Questionnaire. Responses are scored on

the scale 1/Not at all confident = 1 point to 10/Very Confident = 10 points.

Variable: JOBSEEK T1 1

<u>Label</u>: Job-Seeking Self Efficacy Score at T1

Type: Numeric; Range = 1 to 10

Algorithm: JOBSEEK\_T1\_1 = MEAN(BSL52a, BSL52b, BSL52c, BSL52d, BSL52e, BSL52f, BSL53a,

BSL53b, BSL53c, BSL53d, BSL53e, BSL53f)

If all responses are missing, then JOBSEEK\_T1\_1=Missing. Otherwise, calculate the mean

of the non-missing responses.

#### 1.3.2. Job Seeking Self-Efficacy Score at Post-Intervention (T2)

Description: Job Seeking Self-Efficacy score at time point T2 (Post-Intervention) is based on 12 items

(13a through 13f and 14a through 14f) from the EVL Questionnaire. Responses are scored on the scale 1/Not at all confident = 1 point to 10/Very Confident = 10 points.

Variable: JOBSEEK\_T2\_1

Label: Job-Seeking Self Efficacy Score at T2

Type: Numeric; Range = 1 to 10

Algorithm: JOBSEEK\_T2\_1 = MEAN (EVL13a, EVL13b, EVL13c, EVL13d, EVL13e, EVL13f, EVL14a,

EVL14b, EVL14c, EVL14d, EVL14e, EVL14f)

If all responses are missing, then JOBSEEK\_T2\_1=Missing. Otherwise, calculate the mean

of the non-missing responses.

# 1.3.3. Job Seeking Self-Efficacy Score at Month 3 Follow-Up (T3)

<u>Description</u>: Job Seeking Self-Efficacy score at time point T3 (Month 3 follow-up) is based on 12 items

(52a through 52f and 53a through 53f) from the EXQ Questionnaire. Responses are scored on the scale 1/Not at all confident = 1 point to 10/Very Confident = 10 points.

Variable: JOBSEEK\_T3\_1

<u>Label</u>: Job-Seeking Self Efficacy Score at T3

Type: Numeric; Range = 1 to 10

Algorithm: JOBSEEK\_T3\_1 = MEAN (EXQ52a, EXQ52b, EXQ52c, EXQ52d, EXQ52e, EXQ52f, EXQ53a,

EXQ53b, EXQ53c, EXQ53d, EXQ53e, EXQ53f)

If all responses are missing, then JOBSEEK\_T3\_1=Missing. Otherwise, calculate the mean

ofnon-missing responses

## 1.3.4. Change in Job Seeking Self-Efficacy Score from Baseline to Month 3 Follow-Up (T1T3)

<u>Description</u>: Difference between Job Seeking Self-Efficacy score at the Month 3 follow-up (T3) and

the score at Baseline (T1). If the Job Seeking Self-Efficacy score is missing at T3, then the

score from T2 is used to compute the change in score from T1.

Variable: JOBSEEK\_T1T3\_1

Label: Change in Job-Seeking Self Efficacy Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -9 to 9

Algorithm: If JOBSEEK\_T3\_1 not . then JOBSEEK\_T1T3\_1=JOBSEEK\_T3\_1 – JOBSEEK\_T1\_1

Else if JOBSEEK\_T3\_1=. then JOBSEEK\_T1T3\_1=JOBSEEK\_T2\_1 – JOBSEEK\_T1\_1

If JOBSEEK\_T1\_1 is missing, then JOBSEEK\_T1T3\_1=Missing. If JOBSEEK\_T2\_1 and

JOBSEEK T3 1 are missing, then JOBSEEK T1T3 1=Missing.

# 1.4. PROTEAN CAREER ATTITUDES SCALE (PCA) SCORE:

Protean career attitudes are defined as having self-direction in the pursuit of success in one's work. The scale (and the two sub scales) were measured at Baseline (T1) and the Month 3 follow-up (T3). Higher values indicate better attitudes.

# 1.4.1. PCA Subscale 1: Self-Directed Attitudes (SDA) Scale Score

## 1.4.1.1. Self-Directed Attitudes Score at Baseline (T1)

<u>Description</u>: Self-directed Attitudes Scale Score at time point T1 (Baseline) is based on four items

(75b, 75c, 75d, and 76a) from the BSL Questionnaire. Responses are scored as

1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3

points, 4/Agree = 4 points, and 5/Strongly Agree = 5 points.

Variable: SDA\_T1\_1

Label: Self-Directed Attitudes Scale Score at T1

<u>Type</u>: Numeric; Range = 1 to 5

Algorithm: SDA\_T1\_1 = MEAN (BSL75b, BSL75c, BSL 75d, BSL76a)

If all responses are missing, then SDA\_T1\_1=Missing. Otherwise, calculate the mean of

non-missing responses.

# 1.4.1.2. Self-Directed Attitudes Score at Month 3 Follow-Up (T3)

<u>Description</u>: Self-directed Attitudes Scale Score at time point T3 (Month 3 follow-up) is based on four

items (75b, 75c, 75d, and 76a) from the EXQ Questionnaire. Responses are recorded as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3

points, 4/Agree = 4 points, and 5/Strongly Agree = 5 points.

Variable: SDA T3 1

Label: Self-Directed Attitudes Scale Score at T3

Type: Numeric; Range = 1 to 5

<u>Algorithm</u>: SDA\_T3\_1 = MEAN (EXQ75b, EXQ75c, EXQ75d, EXQ76a)

If all responses are missing, then SDA\_T3\_1=Missing. Otherwise, calculate the mean of

non-missing responses.

# 1.4.1.3. Change in Self-Directed Attitudes Score from Baseline to Month 3 Follow-Up (T1T3)

Description: Difference between Self-Directed Attitudes score at time point T3 (Month 3 follow-up)

and time point T1 (Baseline)

Variable: SDA\_T1T3\_1

Label: Change in Self-Directed Attitudes Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -4 to 4

Algorithm:  $SDA_T1T3_1 = SDA_T3_1 - SDA_T1_1$ 

If SDA score at either time point is missing, then SDA T1T3 1=Missing.

# 1.4.2. PCA Subscale 2: Values-Driven Attitudes Scale Score

# 1.4.2.1. Values-Driven Attitudes (VDA) Score at Baseline (T1)

Description: Values driven Attitudes Scale Score at time point T1 (Baseline) is based on 3 items (76b,

76c, and 76d) from the BSL Questionnaire. Response are scored as 1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3 points, 4/Agree = 4

points, and 5/Strongly Agree = 5 points.

Variable: VDA\_T1\_1

<u>Label</u>: Values-Driven Attitudes Scale Score at T1

Type: Numeric; Range = 1 to 5

<u>Algorithm</u>: VDA\_T1\_1 = MEAN (BSL76b, BSL76c, BSL76d)

If all responses are missing, then VDA\_T1\_1=Missing. Otherwise, calculate the mean

ofnon-missing responses.

## 1.4.2.2. Values-Driven Attitudes (VDA) Score at Month 3 Follow-Up (T3)

Description: Values driven Attitudes Scale Score at time point T3 (Month 3 follow-up) is based on 3

items (76b, 76c, and 76d) from the EXQ Questionnaire. Responses are scored as

1/Strongly Disagree = 1 point, 2/Disagree = 2 points, 3/Neither Disagree nor Agree = 3

points, 4/Agree = 4 points, and 5/Strongly Agree = 5 points

Variable: VDA T3 1

<u>Label</u>: Values-Driven Attitudes Scale Score at T3

Type: Numeric; Range = 1 to 5

<u>Algorithm</u>: VDA\_T3\_1 = MEAN (EXQ76b, EXQ76c, EXQ76d)

If all responses are missing, then VDA\_T3\_1=Missing. Otherwise, calculate the mean

ofnon-missing responses.

# 1.4.2.3. Change in Values-Driven Attitudes (VDA) Score from Baseline to Month 3 Follow-Up (T1T3)

<u>Description</u>: Difference between Values-Driven Attitudes Score at time point T3 (Month 3 follow-up)

from time point T1 (Baseline)

Variable: VDA\_T1T3\_1

<u>Label</u>: Change in Values Driven Attitudes Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -4 to 4

Algorithm:  $VDA_T1T3_1 = VDA_T3_1 - VDA_T1_1$ 

If VDA score at either time point is missing, then VDA\_T1T3\_1=Missing.

# 1.4.3. Scale: Protean Career Attitudes (PCA) Scale

# 1.4.3.1. Protean Career Attitudes (PCA) Score at Baseline (T1)

<u>Description</u>: The Protean Career Attitudes Score at T1 is obtained by adding the two subscale scores

defined above: SDA Score at T1 and VDA Score at T1.

Variable: PCA\_T1\_1

Label: Protean Career Attitudes Score at T1

Type: Numeric; Range = 1 to 5

Algorithm:  $PCA_T1_1 = MEAN (SDA_T1_1, VDA_T1_1)$ 

If either SDA or VDA score is missing, then PCA\_T1\_1=Missing.

# 1.4.3.2. Protean Career Attitudes (PCA) Score at Month 3 Follow-Up (T3)

<u>Description</u>: The Protean Career Attitudes Score at T3 is obtained by adding the two subscale scores

defined above: SDA Score at T3 and VDA Score at T3.

Variable: PCA\_T3\_1

Label: Protean Career Attitudes Score at T3

Type: Numeric; Range = 1 to 5

Algorithm: PCA\_T3\_1 = MEAN (SDA\_T3\_1, VDA\_T3\_1)

If either SDA or VDA score is missing, then PCA\_T3\_1=Missing.

# 1.4.3.3. Change in Protean Career Attitudes (PCA) Score from Baseline to Month 3 Follow-Up (T1T3)

<u>Description</u>: Difference between protean career attitudes score at time point T3 (Month 3 follow-up)

and time point T1 (Baseline)

Variable: PCA\_T1T3\_1

<u>Label</u>: Change in Protean Career Attitudes Score from T1 to T3 (T3-T1)

Type: Numeric; Range = -4 to 4

Algorithm:  $PCA_T1T3_1 = PCA_T3_1 - PCA_T1_1$ .

If PCA score at either time point is missing, then PCA\_T1T3\_1=Missing.

# 2. SECONDARY OUTCOMES

#### 2.1. SELF-REPORTED EMPLOYMENT

The primary employment outcome is based on the change in the number of self-report hours worked per week from T1 to T3.

# 2.1.1. Change in Self-Reported Hours Worked Per Week from Baseline to Month 3 Follow-Up (T1T3)

<u>Description</u>: Change in hours worked per week from Baseline to Month 3 follow-up (T1 to T3)

Variable: EMPHOUR\_T1T3\_1

Label: Change in Hours Worked per Week from T1 to T3 (T3-T1)

Type: Numeric; Range = -99 to 99

Algorithm: If BSL9 = 0 then BSL27 = 0

If EXQ9 = 0 then EXQ27 = 0

 $EMPHOUR_T1T3_1 = EXQ27 - BSL27$ 

If hours work per week at either time point is missing, then EMPHOUR\_T1T3\_1=Missing.

# 2.2. SELF-REPORTED SEXUAL RISK BEHAVIORS

## 2.2.1. Self-Reported Sexual Risk Behavior at Baseline (T1)

Description: Sexual Risk behavior is measured using items 239 through 244 from the BSL

Questionnaire. Responses for each question are either Yes (1), No (0) or Missing (.). Risk

Behavior is defined as the mean of responses to the risk behavior questions.

Variable: RISK\_T1\_1

Label: Self-Reported Sexual Risk Behavior at T1

Type: Numeric; Range = 0 to 1

Algorithm:  $RISK_T1_1 = MEAN (BSL239, BSL240, BSL241, BSL242, BSL243, BSL244)$ 

If responses for four or more individual risk behavior questions are missing, then RISK\_T1\_1 = Missing. Otherwise, calculate the mean of non-missing responses.

# 2.2.2. Self-Reported Sexual Risk Behavior at Baseline (T3)

<u>Description</u>: Sexual Risk behavior is measured using items 239 through 244 from the EXQ

Questionnaire. Responses for each question are either Yes (1), No (0) or Missing (.). Risk

Behavior is as the mean of responses to the risk behavior questions.

Variable: RISK\_T3\_1

Label: Self-Reported Sexual Risk Behavior at T3

Type: Numeric; Range = 0 to 1

Algorithm: RISK\_T3\_1 = MEAN (EXQ239, EXQ240, EXQ241, EXQ242, EXQ243, EXQ244)

If responses for four or more individual risk behavior questions are missing, then RISK\_T3\_1 = Missing. Otherwise, calculate the mean of non-missing responses.

# 2.2.3. Change in Self-Reported Risk Behavior from Baseline to Month 3 Follow-Up (T1T3)

Description: Change in Self-Reported Risk Behavior of a participant from Baseline to month 3 follow-

up (T1 to T3)

Variable: RISK\_T1T3\_1

<u>Label</u>: Change in Self-Reported Sexual Risk Behavior from T1 to T3 (T3-T1)

Type: Numeric; Range = -1 to 1

Algorithm: RISK T1T3 1 = RISK T3 1 - RISK T1 1.

If risk behavior at either time point is missing, then RISK\_T1T3\_1 = Missing.

#### 2.3. CHLAMYDIA INFECTIONS:

Chlamydia will be assessed at T1 (Baseline) and T3 (3-month follow-up) using urine, anal, and oral sample tests.

# 2.3.1. Chlamydia Result at Baseline (T1)

## 2.3.1.1. Chlamydia Result based on Oral Sample at T1

<u>Description</u>: The oral sample collection status is recorded in item 10a of the Biospecimen Collection

(BIC1) form and the oral swab Chlamydia result is recorded in item 1a of the

Biospecimen Results (BLR1) Form for Baseline (T1).

Variable: CH\_ORAL\_T1\_1

Label: Assessment of Chlamydia using an Oral Test at T1

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC10a = 1 then CH ORAL T1 1 = [BLR1] BLR1a

Else if [BIC1] BIC10a=1 and [BLR1] BLR1a=. then CH\_ORAL\_T1\_1 = .U

Else if [BIC1] BIC10a=0 then CH\_ORAL\_T1\_1 = .N Else if [BIC1] BIC10a=9 then CH\_ORAL\_T1\_1 = .R Else if [BIC1] BIC10a=. then CH\_ORAL\_T1\_1 = .

# 2.3.1.2. Chlamydia Result based on Anal Sample at T1

Description: The anal sample collection status is recorded in item 11a of the BIC1 form and the anal

swab Chlamydia result is recorded in item 2a of the BLR1 Form for Baseline (T1).

Variable: CH\_ANAL\_T1\_1

<u>Label</u>: Assessment of Chlamydia using an Anal Test at T1

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC11a = 1 then CH\_ANAL\_T1\_1 = [BLR1] BLR2a

Else if [BIC1] BIC11a=1 and [BLR1] BLR2a=. then CH\_ANAL\_T1\_1 = .U

Else if [BIC1] BIC11a=0 then ANAL\_CH\_T1\_1 = .N Else if [BIC1] BIC11a=9 then ANAL\_CH\_T1\_1 = .R Else if [BIC1] BIC11a=. then ANAL\_CH\_T1\_1 = .

# 2.3.1.3. Chlamydia Result based on Urine Sample at T1

<u>Description</u>: The urine sample collection status is recorded in item 12a of BIC1 form and the urine

Chlamydia result is recorded in item 3a of BLR1 Form for Baseline (T1).

<u>Variable</u>: CH\_URINE\_T1\_1

Label: Assessment of Chlamydia using a Urine Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC12a = 1 then CH\_URINE\_T1\_1 = [BLR1] BLR3a

Else if [BIC1] BIC12a=1 and [BLR1] BLR3a=. then CH\_URINE\_T1\_1 = .U

Else if [BIC1] BIC12a=0 then CH\_URINE\_T1\_1 = .N Else if [BIC1] BIC12a=9 then CH\_URINE\_T1\_1 = .R Else if [BIC1] BIC12a=. then CH\_URINE\_T1\_1 = .

# 2.3.2. Chlamydia Result at Month 3 Follow-Up (T3)

# 2.3.2.1. Chlamydia Result based on Oral Sample at T3

<u>Description</u>: The oral sample collection status is recorded in item 10a of the Biospecimen Collection

(BIC2) form and the oral swab Chlamydia result is recorded in item 1a of the

Biospecimen Results (BLR2) Form for 3-Month Follow-up (T3).

Variable: CH\_ORAL\_T3\_1

<u>Label</u>: Assessment of Chlamydia using an Oral Test T3

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC10a = 1 then CH ORAL T3 1 = [BLR2] BLR1a

Else if [BIC2] BIC10a=1 and [BLR2] BLR1a=. then CH\_ORAL\_T3\_1 = .U

Else if [BIC2] BIC10a=0 then CH\_ORAL\_T3\_1 = .N Else if [BIC2] BIC10a=9 then CH\_ORAL\_T3\_1 = .R Else if [BIC2] BIC10a=. then CH\_ORAL\_T3\_1 = .

# 2.3.2.2. Chlamydia Result based on Anal Sample at T3

Description: The anal sample collection status is recorded in item 11a of the BIC2 form and the anal

swab Chlamydia result is recorded in item 2a of the BLR2 Form for the Month 3 follow-

up (T3).

<u>Variable</u>: CH\_ANAL\_T3\_1

Label: Assessment of Chlamydia using an Anal Test T3

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC11a = 1 then CH\_ANAL\_T3\_1 = [BLR2] BLR2a

Else if [BIC2] BIC11a=1 and [BLR2] BLR2a=. then CH\_ANAL\_T3\_1 = .U

Else if [BIC2] BIC11a=0 then CH\_ANAL\_T3\_1 = .N Else if [BIC2] BIC11a=9 then CH\_ANAL\_T3\_1 = .R Else if [BIC2] BIC11a=. then CH\_ANAL\_T3\_1 = .

# 2.3.2.3. Chlamydia Result based on Urine Sample at T3

<u>Description</u>: The urine sample collection status is recorded in item 12a of BIC2 form and the urine

Chlamydia result is recorded in item 3a of BLR2 Form for Month 3 follow-up (T3).

<u>Variable</u>: CH\_URINE\_T3\_1

Label: Assessment of Chlamydia using a Urine Test T3

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC12a = 1 then CH\_URINE\_T3\_1 = [BLR2] BLR3a

Else if [BIC2] BIC12a=1 and [BLR2] BLR3a=. then CH\_URINE\_T3\_1 = .U

Else if [BIC2] BIC12a=0 then CH\_URINE\_T3\_1 = .N Else if [BIC2] BIC12a=9 then CH\_URINE\_T3\_1 = .R Else if [BIC2] BIC12a=. then CH\_URINE\_T3\_1 = .

# 2.3.3. Change in Chlamydia Result from Baseline to Month 3 Follow-Up (T1T3)

# 2.3.3.1. Change in Chlamydia Result based on Oral Samples at T1T3

Description: Change in Chlamydia oral sample result of a participant from Baseline to Month 3

follow-up (T1 to T3)

Variable: CH\_ORAL\_T1T3\_1

Label: Change in Chlamydia Oral Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Oral Result,

-1=Positive to Negative

<u>Algorithm</u>: CH\_ORAL\_T1T3\_1 = CH\_ORAL\_T3\_1 - CH\_ORAL\_T1\_1

If measurement at either time point is missing, then CH ORAL T1T3 1 = missing.

# 2.3.3.2. Change in Chlamydia Result based on Anal Samples at T1T3

Description: Change in Chlamydia anal sample result of a participant from Baseline to Month 3

follow-up (T1 to T3)

Variable: CH\_ANAL\_T1T3\_1

Label: Change in Chlamydia Anal Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Oral Result,

-1=Positive to Negative

Algorithm: CH\_ANAL\_T1T3\_1 = CH\_ANAL\_T3\_1 - CH\_ANAL\_T1\_1

If measurement at either time point is missing, then CH\_ANAL\_T1T3\_1 = missing.

# 2.3.3.3. Change in Chlamydia Result based on Urine Samples at T1T3

Description: Change in Chlamydia urine sample result of a participant from Baseline to Month 3

follow-up (T1 to T3)

Variable: CH\_URINE\_T1T3\_1

Label: Change in Chlamydia Urine Sample Result from T1 to T3 (T3-T1)

Type: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Oral Result,

-1=Positive to Negative

<u>Algorithm</u>: CH\_URINE\_T1T3\_1 = CH\_URINE\_T3\_1 - CH\_URINE\_T1\_1

If measurement at either time point is missing, then CH\_URINE\_T1T3\_1 = missing.

## 2.4. GONORRHEA INFECTIONS:

Gonorrhea will be assessed at T1 (Baseline) and T3 (3-Month follow-up) using urine, anal, and oral sample tests.

## 2.4.1. Gonorrhea Result at Baseline (T1)

# 2.4.1.1. Gonorrhea Result based on Oral Sample at T1

<u>Description</u>: The oral sample collection status is recorded in item 10a of the BIC1 form and the oral

swab Gonorrhea result is recorded in item 1b of the BLR1 Form for Baseline (T1).

Variable: GN\_ORAL\_T1\_1

Label: Assessment of Gonorrhea using an Oral Test at T1

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC10a = 1 then GN\_ORAL\_T1\_1 = [BLR1] BLR1b

Else if [BIC1] BIC10a=1 and [BLR1] BLR1b=. then GN ORAL T1 1 = .U

Else if [BIC1] BIC10a=0 then GN\_ORAL\_T1\_1 = .N Else if [BIC1] BIC10a=9 then GN\_ORAL\_T1\_1 = .R Else if [BIC1] BIC10a=. then GN\_ORAL\_T1\_1 = .

# 2.4.1.2. Gonorrhea Result based on Anal Sample at T1

<u>Description</u>: The anal sample collection status is recorded in item 11a of the BIC1 form and the anal

swab Gonorrhea result is recorded in item 2b of the BLR1 Form for Baseline (T1).

Variable: GN\_ANAL\_T1\_1

Label: Assessment of Gonorrhea using an Anal Test at T1

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC11a = 1 then GN ANAL T1 1 = [BLR1] BLR2b

Else if [BIC1] BIC11a=1 and [BLR1] BLR2b=. then GN\_ANAL\_T1\_1 = .U

Else if [BIC1] BIC11a=0 then GN\_ANAL\_T1\_1 = .N Else if [BIC1] BIC11a=9 then GN\_ANAL\_T1\_1 = .R Else if [BIC1] BIC11a=. then GN\_ANAL\_T1\_1 = .

# 2.4.1.3. Gonorrhea Result based on Urine Sample at T1

<u>Description</u>: The urine sample collection status is recorded in item 12a of BIC1 form and the urine

Gonorrhea result is recorded in item 3b of BLR1 Form for Baseline (T1).

Variable: GN\_URINE\_T1\_1

<u>Label</u>: Assessment of Gonorrhea using a Urine Test at T1

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC1] BIC12a = 1 then GN\_URINE\_T1\_1 = [BLR1] BLR3b

Else if [BIC1] BIC12a=1 and [BLR1] BLR3b=. then GN URINE T1 1 = .U

Else if [BIC1] BIC12a=0 then GN\_URINE\_T1\_1 = .N Else if [BIC1] BIC12a=9 then GN\_URINE\_T1\_1 = .R Else if [BIC1] BIC12a=. then GN\_URINE\_T1\_1 = .

# 2.4.2. Gonorrhea Result at Month 3 Follow-Up (T3)

# 2.4.2.1. Gonorrhea Result based on Oral Sample at T3

<u>Description</u>: The oral sample collection status is recorded in item 10a of the BIC2 form and the oral

swab Gonorrhea result is recorded in item 1b of the BLR2 Form for 3-Month follow-up

(T3).

Variable: GN ORAL T3 1

Label: Assessment of Gonorrhea using an Oral Test T3

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC10a = 1 then GN ORAL T3 1 = [BLR2] BLR1b

Else if [BIC2] BIC10a=1 and [BLR2] BLR1b=. then GN ORAL T3 1 = .U

Else if [BIC2] BIC10a=0 then GN\_ORAL\_T3\_1 = .N Else if [BIC2] BIC10a=9 then GN\_ORAL\_T3\_1 = .R Else if [BIC2] BIC10a=. then GN\_ORAL\_T3\_1 = .

# 2.4.2.2. Gonorrhea Result based on Anal Sample at T3

Description: The anal sample collection status is recorded in item 11a of the BIC2 form and the anal

swab Gonorrhea result is recorded in item 2b of the BLR2 Form for the Month 3 follow-

up (T3).

Variable: GN\_ANAL\_T3\_1

Label: Assessment of Gonorrhea using an Anal Test T3

Type: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC11a = 1 then GN\_ANAL\_T3\_1 = [BLR2] BLR2b

Else if [BIC2] BIC11a=1 and [BLR2] BLR2b=. then GN\_ANAL\_T3\_1 = .U

Else if [BIC2] BIC11a=0 then GN\_ANAL\_T3\_1 = .N Else if [BIC2] BIC11a=9 then GN\_ANAL\_T3\_1 = .R Else if [BIC2] BIC11a=. then GN\_ANAL\_T3\_1 = .

## 2.4.2.3. Gonorrhea Result based on Urine Sample at T3

Description: The urine sample collection status is recorded in item 12a of BIC2 form and the urine

Gonorrhea result is recorded in item 3b of BLR2 Form for Month 3 follow-up (T3).

Variable: GN\_URINE\_T3\_1

Label: Assessment of Gonorrhea using a Urine Test T3

<u>Type</u>: Numeric; Format: 1=Positive, 0=Negative, .U=Unknown, .N=Not Collected, .R=Refused,

.=Missing

Algorithm: If [BIC2] BIC12a = 1 then GN\_URINE\_T3\_1 = [BLR2] BLR3b

Else if [BIC2] BIC12a=1 and [BLR2] BLR3b=. then GN\_URINE\_T3\_1 = .U

Else if [BIC2] BIC12a=0 then GN\_URINE\_T3\_1 = .N

Else if [BIC2] BIC12a=9 then GN\_URINE\_T3\_1 = .R Else if [BIC2] BIC12a=. then GN\_URINE\_T3\_1 = .

# 2.4.3. Change in Gonorrhea Result from Baseline to Month 3 Follow-Up (T1T3)

# 2.4.3.1. Change in Gonorrhea Result based on Oral Samples at T1T3

Description: Change in Gonorrhea oral sample result of a participant from Baseline to Month 3

follow-up (T1 to T3)

Variable: GN\_ORAL\_T1T3\_1

Label: Change in Gonorrhea Oral Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Oral Result, -

1=Positive to Negative

<u>Algorithm</u>: GN\_ORAL\_T1T3\_1 = GN\_ORAL\_T3\_1 - GN\_ORAL\_T1\_1

If measurement at either time point is missing, then GN\_ORAL\_T1T3\_1 = missing.

# 2.4.3.2. Change in Gonorrhea Result based on Anal Samples at T1T3

Description: Change in Gonorrhea anal sample result of a participant from Baseline to Month 3

follow-up (T1 to T3)

Variable: GN\_ANAL\_T1T3\_1

Label: Change in Gonorrhea Anal Sample Result from T1 to T3 (T3-T1)

<u>Type</u>: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea Anal Result, -

1=Positive to Negative

<u>Algorithm:</u> GN\_ANAL\_T1T3\_1 = GN\_ANAL\_T3\_1 - GN\_ANAL\_T1\_1

If measurement at either time point is missing, then GN\_ANAL\_T1T3\_1 = missing.

# 2.4.3.3. Change in Gonorrhea Result based on Urine Samples at T1T3

<u>Description</u>: Change in Gonorrhea urine sample result of a participant from Baseline to Month 3

follow-up (T1 to T3)

Variable: GN URINE T1T3 1

<u>Label</u>: Change in Gonorrhea Urine Sample Result from T1 to T3 (T3-T1)

Type: Numeric; Format: 1=Negative to Positive, 0=No Change in Gonorrhea urine result, -

1=Positive to Negative

<u>Algorithm</u>: GN\_URINE\_T1T3\_1 = GN\_URINE\_T3\_1 - GN\_URINE\_T1\_1

If measurement at either time point is missing, then GN\_URINE\_T1T3\_1 = missing.

## 2.5. REACTIVE HIV TEST

<u>Description</u>: Testing for HIV is conducted at Baseline (T1) and Month 3 follow-up (T3) and indicates

whether or not the test result was reactive or non-reactive. The reactive HIV testing

result for T3 is recorded in item 1a of the BIC2 form.

Variable: HIVREAC\_T3\_1

Label: Reactive HIV Test Result at T3.

<u>Type</u>: Numeric; Format: 0=Non-Reactive, 1=Reactive, .U=Unknown, .N=Not Collected,

.R=Refused, .=Missing

Algorithm: If [BIC2] BIC1=1 then HIVREAC\_T3\_1= [BIC2] BIC1a

Else if [BIC2] BIC1=1 and [BIC2] BIC1a=. then HIVREAC\_T3\_1=.U

Else if [BIC2] BIC1=0 then HIVREAC T3 1 1 = .N

Else if [BIC2] BIC1=9 and [BIC2] BIC1a=9 then HIVREAC\_T3\_1=.R Else if [BIC2] BIC1=. and [BIC2] BIC1a=. then HIVREAC\_T3\_1=.